# 16.1.9 DOCUMENTATION OF STATISTICAL METHODS



## **SAP (PHASE II STUDY)**

EN-SOP-ST-03-Temp-01 V2.0

Version: Final

#### TIRHOL

A Phase 2, Multicenter, Open-Label Study of Tislelizumab (BGB-A317) in

Patients with Relapsed or Refractory Classical Hodgkin Lymphoma

Statistical Analysis Plan

LYSARC: The Lymphoma Academic Research Organisation ☑: Centre Hospitalier Lyon Sud – Bâtiment 2D 69495 Pierre Bénite Cedex - France

Version 1.0 April, 12th 2023

| COORDINATING INVESTIGATOR | |
|------------------------------|--------|
| CO-COORDINATING INVESTIGATOR | |
| COORDINATION CENTER | LYSARC |
| COORDINATION CENTER | LYSARC |

| Initial Version and date of Protocol | v0.0 10JULY2019 |
|--------------------------------------|-----------------|
| Last version and date of Protocol | V5.0 27SEP2022 |
| EudraCT Number | |





## SAP (PHASE II STUDY)

EN-SOP-ST-03-Temp-01 V2.0

Version: Final

## **APPROVAL PAGE**





## SAP (PHASE II STUDY)

EN-SOP-ST-03-Temp-01 V2.0

Version : Final

### **Document History:**

| Version # | Effective Date | Author | Modification Description | Affected |
|-----------|----------------|--------|--------------------------|------------|
| | | | | Paragraphs |
| 1.0 | 12APR2023 | | Document creation | |

## **TABLE OF CONTENTS**

| Li | st of O | utputs | 7 |
|----|----------------|------------------------------------------|----|
| Li | st of Al | bbreviations | 12 |
| 1 | Intro | oduction | 14 |
| 2 | Inve | estigational plan | 15 |
| | 2.1 | Rationale | |
| | 2.2 | Study Design | |
| 3 | | ly objectives and endpoints | |
| | 3.1 | Objectives | |
| | 3.1.1 | • | |
| | 3.1.2 | | |
| | 3.1.3 | Exploratory objectives | 17 |
| | 3.2 | Evaluation endpoints | 17 |
| | 3.2.1 | • | |
| | 3.2.2 | | |
| | 3.2.3 | | |
| | 3.2.4 | | |
| | 3.3 | Follow-up duration | 21 |
| | | • | |
| | 3.4 | Extent of exposure | |
| 4 | Cha | nges from Protocol | 22 |
| 5 | Stat | istical Considerations | 23 |
| | 5.1 | Sample size calculation | 23 |
| | 5.2 | Interim analyses | 23 |
| | 5.3 | Analyses of primary endpoint | 23 |
| | 5.4 | Final analysis | 24 |
| | 5.5 | Analysis Sets | 24 |
| | 5.5.1 | • | |
| | 5.5.2 | | |
| | 5.5.3 | | |
| | F 6 | | |
| | 5.6 | General statistical approach | |
| | 5.6.1<br>5.6.2 | | |
| | 5.6.2 | | |
| | 5.7 | Handling of missing or off-schedule data | |
| | 5.8 | Software | |
| 6 | Ana | lysis Plan | 27 |
| | 6.1 | Study Summary | 27 |
| | 6.1.1 | Overall description | 27 |
| | 6.1.2 | Study dates | 27 |
| | 6.1.3 | Follow-up duration | 27 |
| | 6.2 | Study patients | 27 |
| | | • • | |

| 6.2.1 | Disposition of patients | 27 |
|---|---|---|
| 6.2.2 | Analysis Sets | 27 |
| 6.2.3 | Analysis subsets | 27 |
| 6.3 | Inclusion / Exclusion criteria | 28 |
| 6.4 | Protocol deviations | 28 |
| 6.4.1 | Major protocol deviations | 28 |
| 6.5 | Demographic and other baseline characteristics | 29 |
| 6.6 | Evaluation during study | <b>2</b> 9 |
| 6.6.1 | Clinical examination | 29 |
| 6.6.2 | Tumor assessment | 29 |
| 6.7 | Efficacy Analysis | 30 |
| 6.7.1 | | |
| 6.7.2 | | |
| 6.7.3 | | |
| 6.7.4 | Progression / Relapse | 31 |
| 6.7.5 | New anti-cancer therapy given prior to disease progression | 31 |
| 6.8 | Extent of exposure | 32 |
| 6.8.1 | Cycles | 32 |
| 6.8.2 | Dose | 32 |
| 6.8.3 | Dose modifications | 32 |
| 6.9 | Safety analysis | 32 |
| 6.9.1 | Treatment Emergent Adverse Events | 32 |
| 6.9.2 | Serious Adverse Events | 33 |
| 6.9.3 | Secondary primary malignancies | 33 |
| 6.9.4 | Deaths | 33 |
| 6.9.5 | Clinical Laboratory / Vital signs | 33 |
| 6.9.6 | Pregnancies | |
| 6.10 | Concomitant treatments | |
| 6.10. | 1 Prior treatment reported at enrollment | 34 |
| 6.10. | 2 Concomitant treatments | |
| 7 Stati | istical outputs | 35 |
| 7.1 | Study Summary | 36 |
| 7.1.1 | | |
| 7.1.2 | • | |
| 7.1.3 | • | |
| 7.2 | Study patients | 37 |
| 7.2.1 | ••• | |
| 7.2.2 | | |
| 7.2.3 | • | |
| 7.3 | Inclusion / Exclusion criteria | 41 |
| | Major protocol deviations | |
| | Demographic and other baseline characteristics | |
| 7.5.1 | 0 -1 | |
| 7.5.2 | | |
| 7.5.3<br>7.5.4 | | |
| 7.5.4<br>7.5.5 | | |
| 7.5.6 | · | |
| 7.5.0 | Other chilical examp | |

| 7.6 | Evaluation during study | 60 |
|-------|------------------------------------------------------------|-----|
| 7.6.1 | Clinical examination | 60 |
| 7.6.2 | Tumor assessment | 62 |
| 7.7 | Efficacy Analysis | 70 |
| 7.7.1 | Primary efficacy endpoint analyses | 70 |
| 7.7.2 | Secondary efficacy endpoint analyses | 73 |
| 7.7.3 | Exploratory endpoint analyses | 78 |
| 7.7.4 | Progression / Relapse | 82 |
| 7.7.5 | New anti-cancer therapy given prior to disease progression | 85 |
| 7.8 | Extent of exposure | 87 |
| 7.8.1 | Cycles | 87 |
| 7.8.2 | Pose | 88 |
| 7.8.3 | Dose modifications | 89 |
| 7.9 | Safety analysis | 92 |
| 7.9.1 | Treatment Emergent Adverse Events | 92 |
| 7.9.2 | Serious Adverse Events | 102 |
| 7.9.3 | Second primary malignancies | 106 |
| 7.9.4 | Deaths | 106 |
| 7.9.5 | Clinical Laboratory / Vital signs | 108 |
| 7.9.6 | Pregnancies | 112 |
| 7.10 | Prior and concomitant treatments | 113 |
| 7.10. | 1 Prior treatments reported at enrollment | 113 |
| 7.10. | 2 Concomitant treatments | 113 |

## **LIST OF OUTPUTS**

| Index of tables | |
|---|---|
| Table 5.3-1 Content of analyses for primary endpoint | <b>2</b> 3 |
| Table 5.4-1 Content of final analysis | 24 |
| Table 7.1-1 Number of patients by country and by center – Enrolled set | 36 |
| Table 7.1-2 Number of patients at each timepoint – Safety Analysis set | 36 |
| Table 7.1-3 Inclusion dates - Enrolled sets | 36 |
| Table 7.1-4 Date of last visit last patient - Enrolled set | 36 |
| Table 7.1-5 Follow-up duration - Safety Analysis set | |
| Table 7.2-1 Permanent treatment discontinuation during the study – Safety Analysis set | 37 |
| Table 7.2-2 Patient status - Safety Analysis Set | 38 |
| Table 7.2-3 Patients included in the trial - Enrolled Set | 39 |
| Table 7.2-4 Patients included in the trial with central confirmation of cHL diagnosis - Enrolled Set | 40 |
| Table 7.3-1 Patients with at least one inclusion/exclusion criterion not fulfilled | 44 |
| Table 7.4-1 Major protocol deviations – Enrolled set | 45 |
| Table 7.5-1 Demographic characteristics at inclusion | |
| Table 7.5-2 Histological diagnosis according to local review | |
| Table 7.5-3 Histological diagnosis according to central review | |
| Table 7.5-4 Disease assessments and staging at inclusion | |
| Table 7.5-5 Number of prior lines of therapy for cHL | 48 |
| Table 7.5-6 Overview of nodal/extra-nodal involvement at baseline | |
| Table 7.5-7 Supra-diaphragmatic nodal involvement at baseline | 49 |
| Table 7.5-8 Infra-diaphragmatic nodal involvement at baseline | 49 |
| Table 7.5-9 Other nodal involvement at baseline | |
| Table 7.5-10 Extra-nodal involvement in the Head and Neck Area at baseline | 50 |
| Table 7.5-11 Extra-nodal involvement in Central Nervous System Area at baseline | 50 |
| Table 7.5-12 Extra-nodal involvement in the Digestive Tract Area at baseline | |
| Table 7.5-13 Other extra-nodal involvement at baseline | |
| Table 7.5-14 PET scan at baseline | 54 |
| Table 7.5-15 Sites and methods used for tumor assessment at baseline | 54 |
| Table 7.5-16 Methods of measurements at baseline | 54 |
| Table 7.5-17 Extra-nodal sites evaluable but not measurable at baseline | 55 |
| Table 7.5-18 Medical history | 55 |
| Table 7.5-19 Relevant medical history (including prior cancer) by SOC/PT | 55 |
| Table 7.5-20 Vital signs at baseline | 56 |
| Table 7.5-21 Clinical examination at baseline | 56 |
| Table 7.5-22 Serologies at baseline | 57 |
| Table 7.5-23 Cardiac exam at baseline | 58 |
| Table 7.5-24 Childbearing potential | 58 |
| Table 7.5-25 Pulmonary function test | 59 |
| Table 7.6-1 Clinical examination by cycle during treatment | 60 |
| Table 7.6-2 Performance status (ECOG) by cycle during treatment | 60 |
| Table 7.6-3 Clinical examination by cycle at end of treatment | 60 |
| Table 7.6-4 Performance status (ECOG) by cycle at end of treatment | 61 |
| Table 7.6-5 Clinical examination by cycle during efficacy follow-up | 61 |
| Table 7.6-6 Performance status (ECOG) by cycle during efficacy follow-up | |
| Table 7.6-7 PET scan at each visit during treatment | 62 |
| Table 7.6-8 Sites and methods used for tumor assessment treatment | 63 |
| Table 7.6-9 Methods of measurements during treatment | 64 |
| Table 7.6-10 Extra-nodal sites evaluable but not measurable during treatment | 64 |

| Table 7.6-11 Significant increase in size of non target lesion(s) during treatment | 64 |
|---|---|
| Table 7.6-12 New lymphoma lesion(s) during treatment | 64 |
| Table 7.6-13 Spleen and liver assessment during treatment | 65 |
| Table 7.6-14 Methods of spleen and liver assessment during treatment | 65 |
| Table 7.6-15 Metabolic response during treatment | |
| Table 7.6-16 Radiologic response according to Lugano classification (CT-based) during treatment. | 66 |
| Table 7.6-17 PET scan at each visit at end of treatment | |
| Table 7.6-18 Sites and methods used for tumor assessment treatment at end of treatment | 67 |
| Table 7.6-19 Methods of measurements at end of treatment | 67 |
| Table 7.6-20 Extra-nodal sites evaluable but not measurable at end of treatment | 67 |
| Table 7.6-21 Significant increase in size of non target lesion(s) at end of treatment | |
| Table 7.6-22 New lymphoma lesion(s) at end of treatment | |
| Table 7.6-23 Spleen and liver assessment at end of treatment | |
| Table 7.6-24 Methods of spleen and liver assessment at end of treatment | |
| Table 7.6-25 Metabolic response at end of treatment | |
| Table 7.6-26 Radiologic response according to Lugano classification (CT-based) at end of treatmen | |
| Table 7.6-27 Disease status during efficacy follow-up | |
| Table 7.7-1 ORR* evaluation – Safety Analysis Set | |
| Table 7.7-2 ORR* evaluation – Confirmed cHL Set | |
| Table 7.7-3 ORR* evaluation — Safety Analysis Set | |
| Table 7.7-4 ORR* evaluation — Confirmed cHL Set | |
| Table 7.7-5 CRR evaluation | |
| Table 7.7-6 Events according to Duration of response definitions | |
| Table 7.7-7 Reasons for censoring DOR with censoring on NALT | |
| Table 7.7-8 Duration of response with censoring on NALT —Survival Summary | |
| Table 7.7-9 Duration of response with censoring on NALT — Survival Sammary | |
| Table 7.7-10 Duration of response according to EMA censoring rules – Survival Summary | |
| Table 7.7-11 Duration of response according to EMA censoring rules – Survival Summary | |
| Table 7.7-12 Reasons for censoring DOR with censoring on HSCT | |
| Table 7.7-13 Duration of response with censoring on HSCT —Survival Summary | |
| Table 7.7-14 Duration of response with censoring on HSCT – Survival Stillmary | |
| Table 7.7-15 Time to response | |
| · | |
| Table 7.7-16 Events according to PFS definitions | |
| Table 7.7-17 Reasons for censoring PFS with censoring on NALT | |
| Table 7.7-18 PFS with censoring on NALT – Survival Summary | |
| Table 7.7-19 PFS with censoring on NALT – Survival Estimates | |
| Table 7.7-20 PFS with censoring according to EMA censoring rules – Survival Summary | |
| Table 7.7-21 PFS with censoring according to EMA censoring rules— Survival Estimates | |
| Table 7.7-22 Reasons for censoring PFS with censoring on HSCT | |
| Table 7.7-23 PFS with censoring on HSCT – Survival Summary | |
| Table 7.7-24 PFS with censoring on HSCT — Survival Estimates | |
| Table 7.7-25 Events according to OS definition | |
| Table 7.7-26 OS – Survival Summary | |
| Table 7.7-27 OS – Survival Estimates | |
| Table 7.7-28 Patients presenting with progression/relapse | |
| Table 7.7-29 Progression/relapse documentation | |
| Table 7.7-30 New anti-cancer therapy for progression/relapse | |
| Table 7.7-31 Response after additional treatment(s) | |
| Table 7.7-32 New anti-cancer therapy given prior to progression/relapse | |
| Table 7.8-1 Treatment durations | |
| Table 7.8-2 Tislelizumab cycles administered | |
| Table 7.8-3 Tislelizumah exposure | 88 |

| Table 7.8-4 Modifications of scheduled Tislelizumab infusion by patient | 89 |
|---|---|
| Table 7.8-5 Modifications of scheduled Tislelizumab infusion by modification | 89 |
| Table 7.8-6 Modifications of scheduled Tislelizumab infusion by cycle in cohort 1 | 90 |
| Table 7.8-7 Modifications of scheduled Tislelizumab infusion by cycle in cohort 2 | 90 |
| Table 7.9-1 Overview of Treatment Emergent Adverse Events | 92 |
| Table 7.9-2 Characteristics of Treatment Emergent Adverse Events | |
| Table 7.9-3 Description of TEAEs by SOC/PT | |
| Table 7.9-4 Description of TEAEs by highest grade and SOC/PT - Cohort 1 | |
| Table 7.9-5 Description of TEAEs by highest grade and SOC/PT - Cohort 2 | |
| Table 7.9-6 Description of TEAEs with highest grade >=3 by SOC/PT | |
| Table 7.9-7 Description of treatment-related TEAEs by SOC/PT | |
| Table 7.9-8 Description of treatment-related TEAEs by highest grade and SOC/PT - Cohort 1 | |
| Table 7.9-9 Description of treatment-related TEAEs by highest grade and SOC/PT - Cohort 2 | |
| Table 7.9-10 Description of treatment-related TEAEs with highest grade >=3 by SOC/PT | |
| Table 7.9-11 Description of TEAEs leading to discontinuation or interruption of Tislelizumab by | |
| 0 | |
| Table 7.9-12 Description of fatalFatal* AEs by SOC/PT | |
| Table 7.9-13 Description of infusion-related reaction by PT | |
| Table 7.9-13 Description of severe hypersensitivity reactions and flu-like symptoms by PT | |
| Table 7.9-13 Description of irAE according to investigator by PT | |
| Table 7.9-14 Description of irAEs with grade >= 3 according to Beigene charter | |
| Table 7.9-15 Characteristics of Treatment Emergent Serious Adverse Events | |
| Table 7.9-16 Description of treatment-emergent SAEs by SOC/PT | |
| Table 7.9-17 Description of treatment-emergent SAEs by highest grade and SOC/PT - Cohort 1 | |
| Table 7.9-18 Description of treatment-emergent SAEs by highest grade and SOC/PT - Cohort 2 | |
| Table 7.9-19 Description of treatment-emergent SAEs leading to discontinuation of Tislelizu | |
| SOC/PT | |
| Table 7.9-20 Description of treatment-emergent SAEs leading to discontinuation of Tisleliza | |
| grade and SOC/PT - Cohort 1 | |
| Table 7.9-21 Description of treatment-emergent SAEs leading to discontinuation of Tisleliza | |
| grade and SOC/PT - Cohort 2 | |
| Table 7.9-22 Description of other primary malignancies* by SOC/PT | |
| Table 7.9-23 Deaths | |
| Table 7.9-24 Disease status at death | |
| Table 7.9-25 Hematology: Shifts from baseline to worst post baseline grade - Cohort 1 | |
| Table 7.9-26 Hematology: Shifts from baseline to worst post baseline grade - Cohort 2 | |
| Table 7.9-27 Hematology: Summary of Increase in 2 or More Grades as Compared with B | |
| Cohort 1 | |
| Table 7.9-28 Hematology: Summary of Increase in 2 or More Grades as Compared with Bo | |
| Cohort 2 | |
| Table 7.9-29 Biochemistry: Shifts from baseline to worst post baseline grade - Cohort 1 | |
| Table 7.9-30 Biochemistry: Shifts from baseline to worst post baseline grade - Cohort 2 | |
| Table 7.9-31 Biochemistry: Summary of Increase in 2 or More Grades as Compared with B | |
| Cohort 1 | |
| Table 7.9-32 Biochemistry: Summary of Increase in 2 or More Grades as Compared with B | |
| Cohort 2 | |
| Table 7.9-33 Vital signs during treatment | |
| Table 7.10-1 Corticosteroids treatments reported at enrollment | |
| Table 7.10-2 Prior treatments reported at enrollment | |
| Table 7.10-3 Concomitant treatments | |

| Index of figures | |
|---|---|
| Figure 6.2-1 Analysis Sets | 27 |
| Figure 7.7-1 Duration of response with censoring on NALT | <b>7</b> 5 |
| Figure 7.7-2 Duration of response according to EMA censoring rules | 75 |
| Figure 7.7-3 Duration of response with censoring on HSCT | 76 |
| Figure 7.7-4 PFS with censoring on NALT | 78 |
| Figure 7.7-5 PFS with censoring according to EMA censoring rules | 79 |
| Figure 7.7-6 PFS with censoring on HSCT | 80 |
| Figure 7.7-7 OS | 81 |
| Index of listings | |
| Listing 7.2-1 Permanent treatment discontinuation - Safety Analysis Set (XX patients) | |
| Listing 7.2-2 Patients excluded from Safety Analysis Set (XX patients) | |
| Listing 7.2-3 Patients excluded from Confirmed cHL Set (XX patients) | |
| Listing 7.3-1 Patients with at least one eligibility criterion not fulfilled - Safety Analysis Set (XX | patients |
| Listing 7.4-1 Patients with at least one major protocol deviation – Enrolled Set (XX patients) | |
| Listing 7.5-1 Patients with other nodal involvement localizations at baseline – Safety Analysis | |
| patients) | |
| Listing 7.5-2 Patients with other extra-nodal involvement localizations at baseline – Safety Ana | |
| (XX patients) | |
| Listing 7.5-3 Relevant medical history (including prior cancer) - Safety Analysis Set (XX patient | |
| Listing 7.5-4 Patients with abnormal clinial exam at baseline – Safety Analysis Set (XX patient | |
| Listing 7.5-5 Patients with abnormal cardiac exam at baseline – Safety Analysis Set (XX patients) | |
| Listing 7.6-1 Patients with abnormal clinial exam due to active lymphoma during treatment | |
| Analysis Set (XX patients) | |
| Listing 7.6-2 Patients with abnormal clinial exam due to active lymphoma at end of treatment | _ |
| Analysis Set (XX patients) | |
| Listing 7.6-3 Patients with abnormal clinial exam due to active lymphoma during efficacy follows: | |
| Safety Analysis Set (XX patients) | |
| Listing 7.7-1 Patients with best response "Not Evaluated" according to Lugano classification | |
| Analysis Set (XX patients) | |
| Listing 7.7-2 Patients with best response "Not Evaluated" according to Lugano classific | |
| Confirmed cHL Set (XX patients) | |
| Listing 7.7-3 Patients with monoclonal antibody therapy as progression/relapse treatment | |
| Analysis Set (XX patients) | |
| Listing 7.7-4 Patients with other immunotherapy as progression/relapse treatment – Safety | |
| Set (XX patients) | |
| Listing 7.7-5 Patients with chemotherapy as progression/relapse treatment – Safety Analysis | • |
| patients) | |
| Listing 7.7-6 Patients with radiotherapy as progression/relapse treatment – Safety Analysis | |
| patients) | |
| Listing 7.7-7 Patients with autologous transplant as progression/relapse treatment – Safety | |
| Set (XX patients) | |
| Listing 7.7-8 Patients with allogenic transplant as progression/relapse treatment – Safety Ana | |
| (XX patients) | |
| Listing 7.7-9 Patients with IMiD agents as progression/relapse treatment – Safety Analysis | • |
| patients) | |
| Listing 7.7-10 Patients with epigenetic modifiers agents as progression/relapse treatment | |
| Analysis Set (XX patients) | X/ |

| Listing 7.7-11 Patients with kinase inhibitor as progression/relapse treatment – Safety An | alysis Set (XX |
|---|---|
| patients) | 84 |
| Listing 7.7-12 Patients with Other anti-cancer therapy as progression/relapse treatm | |
| Analysis Set (XX patients) | |
| Listing 7.7-13 Patients with monoclonal antibody therapy given prior to progression/relap | se treatment |
| - Safety Analysis Set (XX patients) | |
| Listing 7.7-14 Patients with other immunotherapy given prior to progression/relapse | |
| Safety Analysis Set (XX patients) | 86 |
| Listing 7.7-15 Patients with chemotherapy given prior to progression/relapse treatm | ent - Safety |
| Analysis Set (XX patients) | |
| Listing 7.7-16 Patients with radiotherapy given prior to progression/relapse treatments | • |
| Analysis Set (XX patients) | |
| Listing 7.7-17 Patients with autologous transplant given prior to progression/relapse | |
| Safety Analysis Set (XX patients) | 86 |
| Listing 7.7-18 Patients with allogenic transplant given prior to progression/relapse treatment to progression to progression transplant given prior to progression transplant given give | |
| Analysis Set (XX patients) | |
| Listing 7.7-19 Patients with IMiD agents given prior to progression/relapse treatment – Sa | |
| Set (XX patients) | |
| Listing 7.7-20 Patients with epigenetic modifiers agents given prior to progression/relaps | |
| - Safety Analysis Set (XX patients) | |
| Listing 7.7-21 Patients with kinase inhibitor given prior to progression/relapse treatments | |
| Analysis Set (XX patients) | |
| Listing 7.7-22 Patients with Other anti-cancer therapy given prior to progression/relapse | treatment – |
| Safety Analysis Set (XX patients) | |
| Listing 7.8-1 Drug withdrawn due to AE - Safety Analysis Set (XX drug withdrawn rep | |
| patients) | |
| Listing 7.8-2 Drug interrupted due to AE - Safety Analysis Set (XX drug interrupted rep | |
| patients) | |
| Listing 7.8-3 Drug delayed due to AE - Safety Analysis Set (XX drug delayed reported by | |
| Listing 7.9-1 Fatal* AEs - Safety Analysis Set (XX AEs in XX patients) | |
| Listing 7.9-4 All grade immune related Adverse Events according to investigator - Safety | |
| (XX AE reported by XX patients) | 99 |
| Listing 7.9-3 Immune related Adverse Events with grade >=3 - Safety Analysis Set (XX AE | |
| XX patients) | |
| Listing 7.9-4 All grade immune related Adverse Events according to Beigene charter - Sa | |
| Set (XX AE reported by XX patients) | |
| Listing 7.9-5 Treatment-emergent SAEs reported by patients - Safety Analysis Set (XX SAEs | |
| XX patients) | |
| Listing 7.9-6 Narratives of other primary malignancies - Safety Analysis Set (XX other | _ |
| reported by XX patients) | |
| Listing 7.9-7 Deaths - Safety Analysis Set (XX patients) | |
| Listing 7.9-8 Narratives of deaths due to SAE - Safety Analysis Set (XX patients) | |
| Listing 7.9-9 Narratives of pregnancies - Safety Analysis Set (XX patients) | |
| Listing 7.10-1 Concomitant treatments - Safety Analysis Set (XX AEs in XX patients) | 114 |

### **LIST OF ABBREVIATIONS**

AE Adverse Event

AESI Adverse Event of Specific Interest

ALT alanine aminotransferase
AST aspartate aminotransferase
cHL classical Hodgkin lymphoma

CI Confidence Interval
CNS Central Nervous System
CR Complete Response
CT Computed Tomography

CTCAE Common Terminology Criteria for Adverse Events

ECG electrocardiogram

ECOG Eastern Cooperative Oncology Group

EoT End of Treatment

ESR Erythrocyte Sedimentation Rate

FDG fluorodeoxyglucose

FFPE formalin-fixed, paraffin-embedded

HBc hepatitis B core HBs hepatitis B surface

HBs Ag hepatitis B surface antigen

HBV Hepatitis B virus HCV Hepatitis C virus

HIV Human immunodeficiency virus

HSCT Hematopoietic Stem Cell Transplantation

IR indeterminate response irAE Immune-related Adverse Event

LDi longest transverse diameter of a lesion

LYRIC Lymphom Response to Immunomodulatory Therapy Criteria

MRI Magnetic Resonance Imaging
MRT Magnetic Resonance Tomography

NCI National Cancer Institute

NMR Nuclear Magnetic Resonance Imaging

ORR Overall response Rate
OS Overall Survival
PD Progressive Disease
PD-1 programmed cell death-1

PD-L1 programmed death ligand-1, programmed death receptor ligand-1,

programmed death-1 ligand-1

PET 18F-FDG Positron Emission Tomography

PFS Progression Free Survival

PK Pharmacokinetics

PPD product of the LDi and perpendicular diameter

PT Preferred Term
QoL Quality Of Life

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SMC Safety Monitoring Comittee

SOC System Organ Class
SPD Sum of Product Diameters

TEAE Treatment Emergent Adverse Event

ULN

Upper Limit of Normal

Page 14

### 1 Introduction

This document describes the statistical analyses and the different layouts for tables and listings to be produced for the protocol TIRHOL titled "A Phase 2, Multicenter, Open-Label Study of Tislelizumab (BGB-A317) in Patients with Relapsed or Refractory Classical Hodgkin Lymphoma". Interim safety review is presented in the Safety Monitoring Committee (SMC) charter.

The statistical analysis plan (SAP) provides a comprehensive and detailed description of the strategy, rationale, and statistical methods to be applied to assess the efficacy and safety of tislelizumab in patients with relapse or refractory classical Hodgkin Lymphoma (cHL).

The purpose of the SAP is to ensure the credibility of the study findings by pre-specifying the statistical approaches before database lock. Data will be regularly reviewed by the Safety Monitoring Committee (SMC) and Sponsor personnel.

The SAP is finalized and signed prior to the clinical database lock.

#### 2 **INVESTIGATIONAL PLAN**

#### 2.1 Rationale

PD-L1 overexpression in HL cells may indicate a genetically determined vulnerability of lymphoma cells to PD-1 blockade. Furthermore, clinical data from other PD-1 inhibitors, nivolumab and pembrolizumab, in cHL, coupled with early data of tislelizumab in Chinese patients with cHL, support the rationale to further explore tislelizumab in a broader population of patients with cHL.

The rationale for this study is further supported by in vivo tumor growth inhibition studies, which demonstrated that tislelizumab has significantly higher anti-tumor activities than nivolumab or pembrolizumab in mouse models carrying allogenic human cancer cells and peripheral blood mononuclear cells (BeiGene internal data).

The efficacy of tislelizumab has also been demonstrated in 70 Chinese patients with cHL. In these patients treated with tislelizumab monotherapy, the ORR was 85.7%, with a CR rate of 61.4%. Tislelizumab was generally well tolerated. The reported ORR and CR rates are higher than those observed with other PD-1 inhibitors. Therefore, study of this molecule in a global setting is warranted. In light of these preliminary safety and efficacy results for monotherapy tislelizumab, coupled with the finding that patients' body weight is not a significant covariate in the clearance of tislelizumab, a fixed dose of tislelizumab at 200 mg once every 3 weeks will be explored in this study.

### 2.2 Study Design

This is a Phase 2, multicenter, open-label study of tislelizumab in patients with relapsed/refractory cHL. The primary efficacy endpoint is overall response rate (ORR), defined as the proportion of patients who achieve a best response of complete response (CR) or partial response (PR), as determined by the investigator per the Lugano Classification.

Approximately 42 patients with relapsed/refractory cHL will be enrolled into one of two cohorts based on prior therapies received: Cohort 1 will include patients who have failed to achieve a response or who have had disease progression after autologous hematopoietic stem cell transplantation (HSCT); Cohort 2 will include patients who have failed to achieve a response or who have had disease progression after at least 1 prior systemic regimen for cHL and are not candidates for autologous or allogeneic HSCT. The primary efficacy analysis will be performed for both cohorts combined, and subgroup analyses by cohorts will be performed.

All patients will receive tislelizumab 200 mg intravenously every 3 weeks until disease progression, unacceptable toxicity, or study withdrawal for other reasons. The end of the study is expected to occur after end of follow-up of last patient. Patients who remain on study treatment at the end of the study may have an opportunity to receive tislelizumab in a separate rollover or extension protocol. A patient in Cohort 2 who achieves a complete remission and is otherwise a candidate for autologous HSCT may proceed to autologous HSCT at the discretion of the investigator and with approval from the sponsor. The investigator should contact the sponsor to discuss autologous HSCT and tislelizumab maintenance therapy post-autologous HSCT.

Treatment with tislelizumab will be open label. Screening procedures must be performed within 28 days prior to the first dose of study treatment, unless noted otherwise. Once all screening assessments have been completed and study eligibility has been confirmed, study treatment must commence within 14 days of confirmation, which is within the 28-day screening window prior to the first dose of study treatment.

#### **Study Assessments**

At screening, written informed consent and medical history will be collected, and eligibility based on inclusion and exclusion criteria will be determined. Baseline assessments will include pulmonary function test, hepatitis B and C serologies (and DNA levels, if necessary), and echocardiogram or

multigated acquisition scan. HIV results will be recorded if previously known. Throughout the study, vital signs, physical examination, Eastern Cooperative Oncology Group (ECOG) performance status, complete blood count with differential, and serum chemistry panel will be monitored. Additional assessments will include height and weight, 12-lead electrocardiogram (ECG), erythrocyte sedimentation rate, pregnancy test (if applicable), and thyroid function evaluation.

Tumor assessments will be performed using PET-CT at screening, at Week 12 from Cycle 1 Day 1, every 12 weeks for 96 weeks, and every 24 weeks (± 14 days) thereafter until disease progression. Computed tomography (CT) with contrast will be performed at screening and every 24 weeks starting from Cycle 1 Day 1 until disease progression. Patient-reported outcomes (European Quality of Life 5-Dimensions 5-Levels health questionnaire [EQ-5D-5L] and European Organisation for Research and Treatment of Cancer Quality of Life cancer core questionnaire [EORTC QLQ-C30]) will also be assessed.

Pharmacokinetic (PK) and immunogenicity analyses will be conducted. For biomarker analyses, blood samples, archival and/or fresh tumor tissue samples will be collected.

Safety assessments will include a review of adverse events (AEs), serious adverse events (SAEs), clinical laboratory tests, physical examinations, pulmonary and cardiac function tests, electrocardiograms, ECOG performance status, and vital signs. All AEs and laboratory safety measurements will be graded per the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0. A safety follow-up visit will be mandatory. All AEs and SAEs occurred within 90 days after the last dose of study treatment, regardless of relationship to study drug, will be reported. A Safety Monitoring Committee will review safety data after at least 20 patients have been on treatment for at least 9 weeks.

### STUDY OBJECTIVES AND ENDPOINTS

### 3.1 Objectives

#### 3.1.1 Primary objective

The primary objective of the study is to evaluate the efficacy of tislelizumab in patients with relapsed/refractory cHL, as measured by the overall response rate (ORR) per the Lugano Classification (Cheson et al 2014) and determined by the investigator.

### 3.1.2 Secondary objectives

The secondary objectives of the study are:

- To evaluate the efficacy of tislelizumab as measured per the Lugano Classification and determined by the investigator for the following:
  - Complete response rate
  - Duration of response
  - Time to response
- To evaluate the safety and tolerability of tislelizumab

### 3.1.3 Exploratory objectives

The exploratory objectives of the study are:

- To evaluate the efficacy of tislelizumab for the following:
  - o Progression-free survival, as measured per the Lugano Classification (Cheson et al 2014) and determined by the investigator
  - o Overall survival

### 3.2 Evaluation endpoints

#### 3.2.1 Primary efficacy endpoint

The ORR is defined as the proportion of patients who achieve a best response of complete response or partial response by positron emission tomography-computed tomography (PET-CT) per the Lugano Classification (Cheson et al 2014) and determined by the investigator (= best overall response).

For each evaluation, the metabolic response (based on PET-CT) is used if available, otherwise the radiological response (based on CT) is used. Best overall response is defined as the best response recorded from the first dose of tislelizumab until data cut-off or the start of a new anti-lymphoma therapy, whichever occurs first. Patients with no post-baseline response assessment (due to any reason) will be considered as non-responders.

Subgroup analyses by cohorts will be performed for best overall response.

#### 3.2.2 Secondary efficacy endpoints

They are assessed by the investigator using the Lugano Classification.

#### 3.2.2.1 Complete response rate

Complete response rate (CRR) is defined as the proportion of patients who achieve a best response of complete response.

Patients with no post-baseline response assessment (due to any reason) will be considered nonresponders.

#### 3.2.2.2 Duration of response

Duration of response is defined as the time from the date that response criteria are first met to the date that disease progression is objectively documented or death, whichever occurs first. For patients with no event, the duration of response is censored at cut-off date or end of study date, whichever occurs first.

Only patients who have achieved an overall response according to primary efficacy endpoint definition will be included in the analysis of duration of response.

Patients who received other new anti-lymphoma therapies (NALT), including HSCT, before having an event (disease progression or death, whichever occurs first), will be censored.

In addition, sensitivity analyses will be performed using the European Medicines Agency (EMA) censoring rules and censoring only for HSCT.

#### Details of censoring rules:

| Situation before the | Censoring "at NALT" | | Censoring "EMA" | | Censoring "only for<br>HSCT" | |
|---|---|---|---|---|---|---|
| date of data cut-off | Date of event or censoring | Censored | Date of event or censoring | Censored | Date of event or censoring | Censore<br>d |
| Death from any cause<br>without prior<br>progression/relapse<br>nor NALT (including<br>HSCT) | Death | No | Death | No | Death | No |
| Death from any cause<br>strictly after NALT but<br>no HSCT started<br>without<br>progression/relapse | Last tumor<br>assessment<br>before NALT | Yes | Death | No | Death | No |
| Death from any cause<br>strictly after HSCT<br>started without<br>progression/relapse | Last tumor<br>assessment<br>before HSCT | Yes | Death | No | Date of the<br>HSCT | Yes |
| Progression/relapse<br>without prior NALT<br>(followed by death or<br>not) | Progression/r<br>elapse | No | Progression/r<br>elapse | No | Progression/r<br>elapse | No |
| Progression/relapse<br>strictly after start of<br>NALT but no HSCT<br>(followed by death or<br>not) | Last tumor<br>assessment<br>before NALT | Yes | Date of<br>progression/r<br>elapse | No | Date of<br>progression/r<br>elapse | No |
| Progression/relapse<br>strictly after HSCT<br>(followed by death or<br>not) | Last tumor<br>assessment<br>before HSCT | Yes | Date of<br>progression/r<br>elapse | No | Date of HSCT | Yes |
| No<br>progression/relapse,<br>nor death, nor NALT | Last tumor<br>assessment*<br>before cut-off | Yes | Last tumor<br>assessment*<br>before cut-off | Yes | Last tumor<br>assessment*<br>before cut-off | Yes |

| No<br>progression/relapse,<br>nor death but start of<br>NALT no HSCT | Last tumor<br>assessment<br>before NALT | Yes | Last tumor<br>assessment*<br>before cut-off | Yes | Last tumor<br>assessment*<br>before cut-off | Yes |
|---|---|---|---|---|---|---|
| No progression/relapse, nor death but HSCT | Last tumor<br>assessment<br>before HSCT | Yes | Last tumor<br>assessment*<br>before cut-off | Yes | Date of HSCT | Yes |
| Lost to follow up with at least one tumor assessment post response | Last tumor<br>assessment*<br>before lost to<br>follow-up | Yes | Last tumor<br>assessment*<br>before lost to<br>follow-up | Yes | Last tumor<br>assessment*<br>before lost to<br>follow-up | Yes |
| Lost to follow up without tumor assessment post response | Date of response | Yes | Date of response | Yes | Date of response | Yes |

<sup>\*</sup> defined as the date of last PET/CT scan

Note: if progression/relapse or death occurs the same day as start of a NALT, event is considered for survival analyses.

#### 3.2.2.3 Time to response

Time to response is defined as the time from the date of the first dose of tislelizumab to the time the response criteria are first met.

Only patients who have achieved an overall response will be included in the analysis of time to response.

### 3.2.3 Secondary safety endpoints

Safety endpoints will include:

- Extent of exposure:
  - o Number of cycles received, duration of exposure, cumulative dose received, dose intensity and relative dose intensity
  - o Dose interruption, modification, or delay, drug discontinuation
- The incidence and severity of adverse events according to NCI-CTCAEv5.0
  - All Treatment Emergent Adverse Event (TEAE)
  - Immune-related Adverse Event (irAE)
  - o SAEs
  - Deaths
  - TEAEs with Grade 3 or above
  - Treatment-related TEAEs
  - o Treatment-related TEAEs with Grade 3 or above
  - o TEAEs that led to treatment discontinuation or dose interruption
- Changes in vital signs:
  - o descriptive summary by visit
- **Physical findings**
- Clinical laboratory results:
  - o descriptive summary and their changes from baseline

Graphical displays may be provided where useful to assist in the interpretation of results

### 3.2.4 Exploratory endpoints

### 3.2.4.1 Progression-free survival

Progression-free survival is as assessed by the investigator using the Lugano Classification and defined as the time from the first dose of tislelizumab to the date of disease progression or death, whichever occurs first.

Patients who receive other anticancer therapies, including HSCT (in Cohort 2), before having an event (disease progression or death, whichever occurs first), will be censored.

In addition, sensitivity analyses will be performed using EMA censoring rules and censoring only for HSCT.

### Details of censoring rules:

| City at least and the | Censoring "a | t NALT" | Censoring "EMA" | | Censoring "only for HSCT | |
|---|---|---|---|---|---|---|
| Situation before the date of data cut-off | Date of event | Censored | Date of event | Censored | Date of event | Censore |
| | or censoring | | or censoring | | or censoring | d |
| Death from any cause without prior progression/relapse nor NALT (including HSCT) | Death | No | Death | No | Death | No |
| Death from any cause<br>strictly after NALT but<br>no HSCT started<br>without<br>progression/relapse | Start of the<br>NALT | Yes | Death | No | Death | No |
| Death from any cause<br>strictly after HSCT<br>started without<br>progression/relapse | Date of the<br>HSCT | Yes | Death | No | Date of the<br>HSCT | Yes |
| Progression/relapse<br>without prior NALT<br>(followed by death or<br>not) | Progression/r<br>elapse | No | Progression/r<br>elapse | No | Progression/r<br>elapse | No |
| Progression/relapse<br>strictly after start of<br>NALT but no HSCT<br>(followed by death or<br>not) | Start of the<br>NALT | Yes | Date of<br>progression/r<br>elapse | No | Date of progression/r elapse | No |
| Progression/relapse<br>strictly after HSCT<br>(followed by death or<br>not) | Date of HSCT | Yes | Date of progression/r elapse | No | Date of HSCT | Yes |
| No<br>progression/relapse,<br>nor death, nor NALT | Last tumor<br>assessment*<br>before cut-off | Yes | Last tumor<br>assessment*<br>before cut-off | Yes | Last tumor<br>assessment*<br>before cut-off | Yes |
| No<br>progression/relapse,<br>nor death but start of<br>NALT no HSCT | Start of the<br>NALT | Yes | Last tumor<br>assessment*<br>before cut-off | Yes | Last tumor<br>assessment*<br>before cut-off | Yes |

/

| No<br>progression/relapse,<br>nor death but HSCT | Date of HSCT | Yes | Last tumor<br>assessment*<br>before cut-off | Yes | Date of HSCT | Yes |
|---|---|---|---|---|---|---|
| Lost to follow up with at least one tumor assessment post baseline | Last tumor<br>assessment*<br>before lost to<br>follow-up | Yes | Last tumor<br>assessment*<br>before lost to<br>follow-up | Yes | Last tumor<br>assessment*<br>before lost to<br>follow-up | Yes |
| Lost to follow up<br>without tumor<br>assessment post<br>baseline | Date of first<br>dose | Yes | Date of first<br>dose | Yes | Date of first<br>dose | Yes |

<sup>\*\*</sup> defined as the date of last PET/CT scan

Note: if progression/relapse or death occurs the same day as start of a NALT, event is considered for survival analyses.

#### 3.2.4.2 Overall survival

Overall survival is defined as the time from the first dose of tislelizumab to the date of death from any cause.

Overall survival will be censored at the last date known to be alive for patients alive at cut-off date. Last date known to be alive is last contact date (max of any exam, any treatment intake, progression, AE,EOS).

Censoring rules used for the OS analysis:

| Situation | Date of event or Censoring | Outcome |
|---|---|---|
| Death from any cause | Date of death | Event |
| Patients with no post-baseline information | Date of first dose | Censored |
| Patient alive | Date of last known alive | Censored |
| Lost to follow-up | Date of last known alive | Censored |

Note: A contact can just be phone call

### 3.3 Follow-up duration

The follow-up duration is defined as the time between the date of the the first dose of tislelizumab and the last contact date (max of any exam, any treatment intake, progression, AE,EOS). Deceased patients are censored at the date of death.

### 3.4 Extent of exposure

- Duration of treatment:

The duration of Tislelizumab treatment (weeks) is calculated as (date of last dose + 21 days - date of first dose)/7.

- Cycles administered
- Cumulative total dose
- Dose intensity:

The dose intensity is defined as: Cumulative total dose received / duration of treatment in days (duration of treatment = date of last dose + 21 days - date of first dose)

Relative dose intensity:

The relative dose intensity is defined as: Dose intensity/Planned dose intensity (Planned dose intensity = 200mg/21 days)

- Modifications of scheduled Tislelizumab infusion

## **4** CHANGES FROM PROTOCOL

No changes from protocol

## STATISTICAL CONSIDERATIONS

### 5.1 Sample size calculation

A total of approximately 42 patients will be enrolled.

The results from a previous clinical trial of tislelizumab (Song et al 2018) yielded an ORR of 85.7% in a predominantly brentuximab vedotin-naive population.

Assuming an alternative ORR of 65% compared to the null ORR of 45% in Cohort 1 and Cohort 2 combined, using a binomial exact test, the power to reject the null hypothesis with 42 patients at a 1sided alpha of 0.05 is greater than 80%.

Power and boundary calculations were performed using East version 6.4.1.

### 5.2 Interim analyses

No interim analysis is planned for this study

### 5.3 Analyses of primary endpoint

One analysis is planned with both cohort combined.

The primary efficacy analysis for both cohorts combined will be conducted at least 12 weeks after the last patient has been dosed, either having undergone the first response assessment or having withdrawn prior to the first response assessment.

All data <= cutoff date will be analyzed, meaning that the data after the cutoff date will be neither analyzed nor displayed in the report.

Table 5.3-1 Content of analyses for primary endpoint

| | Analysis of primary endpoint |
|--------------------------------|------------------------------|
| Study summary | Yes |
| Study patients | Yes |
| Inclusion/exclusion criteria | Yes |
| Major protocol deviation | Yes |
| Demographics and other | Yes |
| baseline characteristics | |
| Evaluation during study | Yes |
| Efficacy analysis | |
| Primary efficacy endpoint | Yes |
| Secondary efficacy endpoints | Yes |
| Exploratory enpoints (PFS, OS) | Yes |
| Other exploratory endpoints | No |
| Progression/Relapse | Yes |
| New anti-cancer therapy given | Yes |
| prior to progression/relapse | |

| Extent of exposure | Yes |
|------------------------|-----|
| Safety analysis | Yes |
| Concomitant treatments | Yes |

### 5.4 Final analysis

An end-of-study analysis will be performed. The end of the study will occur after end of follow-up of last patient.

At that time, all data will be analyzed.

Efficacy analyses will be performed by cohort, and safety analyses will be performed by cohort and overall.

**Table 5.4-1 Content of final analysis** 

| | Final analysis |
|--------------------------------|-------------------------------|
| Study summary | Yes |
| Study patients | Yes |
| Inclusion/exclusion criteria | Yes |
| Major protocol deviation | Yes |
| Demographics and other | Yes |
| baseline characteristics | |
| Evaluation during study | Yes |
| Efficacy analysis | |
| Primary efficacy endpoint | Yes |
| Secondary efficacy endpoints | Yes |
| Exploratory endpoint (PFS, OS) | Yes |
| Other exploratory endpoints | Yes but in separate report(s) |
| Progression/Relapse | Yes |
| New anti-cancer therapy given | Yes |
| prior to progression/relapse | |
| Extent of exposure | Yes |
| Safety analysis | Yes |
| Concomitant treatments | Yes |

## 5.5 Analysis Sets

### 5.5.1 Enrolled Set

The Enrolled Set includes all patients enrolled in the combined cohorts with a signed informed consent.

#### 5.5.2 Safety Analysis Set

The Safety Analysis Set includes all patients who receive at least one dose of tislelizumab. This will be the primary analysis set for the efficacy and safety analyses.

#### 5.5.3 Analysis subsets

The Confirmed cHL Set includes all patients included in the safety analysis set and with a central confirmation of diagnosis.

### 5.6 General statistical approach

### 5.6.1 Statistical analysis

Quantitative variables (including time to response) will be summarized in tables displaying number of observations, mean, standard deviation, median, range; quartiles will also be presented when considered relevant.

Qualitative variables will be expressed as frequencies and percentages (of non-missing data).

**Response** will be described as frequencies and percentages (including missing data).

Response rates will be expressed as percentages with 95% confidence limits according to Exact Pearson-Clopper method. Patients with no post-baseline response assessment (due to any reason) will be considered non-responders.

#### For primary endpoint:

A binomial exact test will be performed to test the null hypothesis (H<sub>0</sub>: ORR = 0.45). If the one-sided pvalue is less than or equal to 0.05 (which is equivalent to observing 25 or more responders out of 42 patients), it will be concluded that single agent tislelizumab statistically significantly increases ORR compared to the historical control.

A two-sided Clopper-Pearson 90% CI will also be constructed to be consistent with the one-sided 0.05 type 1 error.

#### Time to event variables

The median follow-up throughout the study will be calculated using a reverse Kaplan Meier plot of time to death with 95% CIs.

The distribution of DOR, PFS and OS will be estimated using the Kaplan-Meier method.

Median and other quartiles will be estimated with 95% CI using the Brookmeyer and Crowley method (Brookmeyer and Crowley 1982). Survival rate at selected time points will be estimated with its 95% CI using Greenwood's formula.

#### 5.6.2 Statistical methods

Response rates will be estimated with its Pearson-Clopper 95% confidence intervals.

The Kaplan Meier method, also known as the "product-limit method", is a non-paramatric method for estimating the probability of survival at any given point in time. The kaplan-meier method handles both censored and uncensored data.

For survival, medians and quartiles will be estimated with its 95% confidence intervals using Brookmeyer and Crowley method and survival rates will be estimated with their confidence intervals using Greenwood's formula.

#### 5.6.3 Statistical Approach for control of Alpha

No control of alpha is needed.

### 5.7 Handling of missing or off-schedule data

#### Missing data

Incomplete dates for "onset date of AE" and "date when AE became serious" will be imputed as follows:

- If only "day" is missing:
  - If "month/year" is the same as the first intake date of treatment, then "day" will be imputed by the day of first intake if first intake date is non-missing.
  - Otherwise "day" will be imputed by "01".
- If "month" and/or "year" is missing: No imputation will be done.

Note: Chronological order of imputed dates of AE will be checked.

### 5.8 Software

All outputs will be produced using SAS version 9.3 or higher and AdClin version 3.2.2 or higher.

### **6** Analysis Plan

### 6.1 Study Summary

Study Summary will be performed on the Enrolled Set.

#### 6.1.1 Overall description

- Number of patients
- Number of patients by country
- Number of patients by center
- Number of patients at each timepoint (cycle, evaluation, ...)

### 6.1.2 Study dates

- First/Last Date of inclusion
- Date of last Visit Last Patient

### 6.1.3 Follow-up duration

Follow-up duration (figure and table) based on OS follow-up

### 6.2 Study patients

#### 6.2.1 Disposition of patients

Patient disposition will be based on the enrolled set and tabulated for the following categories:

- Number of patients enrolled;
- Number of patients who received at least one dose of Tislelizumab
- Number (percentage) of patients who permanently discontinued treatment;
- If permanent treatment discontinuation, number of last cycle performed
- Reason for treatment discontinuation;
- Patient status (treatment ongoing, efficacy follow up or end of study)

In addition, the listing of patients who permanently discontinued treatment will be displayed with reason.

### 6.2.2 Analysis Sets

Number of patients in each set described in the section §5.5 will be computed. Listing of patients excluded from each set will be displayed with reason

#### Figure 6.2-1 Analysis Sets

### 6.2.3 Analysis subsets

In the event that some patients do not have central confirmation of cHL diagnosis:

Number and percentage of patients in Confirmed cHL Set

### 6.3 Inclusion / Exclusion criteria

Description of the inclusion / exclusion criteria will be performed on the Enrolled set.

The following description will be performed:

- Inclusion criteria
- Exclusion criteria
- Patients with at least one inclusion/exclusion criterion not fulfilled will be presented and listed

### 6.4 Protocol deviations

### 6.4.1 Major protocol deviations

The following description will be performed on the Safety Analysis set:

- Patients with at least one major protocol deviation
- Inclusion/exclusion criterion not fulfilled
- Treatment withdrawal for major protocol devation

Listing of patients with at least one major protocol deviation will be displayed.

Page 29

### 6.5 Demographic and other baseline characteristics

The following items will be described on the Safety Analysis set:

- Demographics
- Disease characteristics
  - o Diagnosis
  - o Disease assessment
  - Previous treatment lines
  - Nodal and extra-nodal involvement
  - PET scan (including bone marrow involvment)
  - Tumor assessement
- Serologies
- Vital signs (see Instruction \$6.9.5)
- Cardiac exams
- Other clinical exams
- Relevant medical history

### 6.6 Evaluation during study

Assessments during treatment and follow-up will be described on safety set.

Two follow-up periods are considered:

Safety follow up: the mandatory Safety Follow-up Visit should be conducted within 30 days (+ 7 days) of the last dose of study treatment.

Efficay follow-up: Following completion of the Safety follow-up phase, every effort should be made to follow patients for survival and for SAEs approximately every 90 days (± 14 days) until PD, withdrawal of consent, death, loss to follow-up, or EOS, whichever occurs first.

#### 6.6.1 Clinical examination

The following items will be described (each cycle during treatment; each visit during efficacy follow-up):

- Results of clinical examination
- Performance status

#### 6.6.2 Tumor assessment

The following items will be described (At Week 12 from C1D1, then every 12 weeks for 96 weeks, and every 24 weeks thereafter, during treatment; every 90 days during efficacy follow-up):

- PET scan and bone marrow involvement
- CT scan
- Sites and methods used for tumor assessment
- Extra-nodal sites but not measurable
- Significant increase in size of non target lesion(s)
- New lymphoma lesion(s) from screening
- Spleen and liver assessment
- Response

### **6.7** Efficacy Analysis

Efficacy analysis will be performed on the Safety Analysis Set according to statistical methods defined in section §5.6.1.

#### 6.7.1 Primary efficacy endpoint analyses

#### 6.7.1.1 Main analysis

The following analyses will be performed:

- Number and percentage of patients falling into each of the response categories
- ORR and its corresponding Clopper-Pearson 95% confidence interval
- Corresponding 90% confidence interval
- Associated binomial test
- Listing of patients with best response Not evaluated

### **6.7.1.2** Sensitivity analysis

In the event that some patients do not have central confirmation of cHL diagnosis, a sensitivity analysis may be performed on the patients in the Safety Analysis Set with central confirmation of cHL diagnosis.

#### 6.7.1.3 Subgroup analyses

Subgroup analyses will be performed by cohort:

- Number and percentage of patients falling into each of the response categories
- ORR and its corresponding Clopper-Pearson 95% confidence interval

### 6.7.2 Secondary efficacy endpoint analyses

#### 6.7.2.1 Complete response rate

The following analyses will be performed:

- Number and percentage of patients falling into each of the response categories
- CRR and its corresponding Clopper-Pearson 95% confidence interval

### **6.7.2.2** Duration of response

The following analyses will be performed:

- Type of event
- Survival curve of duration of response
- Quartiles of survival
- Survival rates at timepoints

#### 6.7.2.3 Time to response

The following analyses will be performed:

Number of observations, mean, standard deviation, median, range, quartiles

### 6.7.3 Exploratory endpoint analyses

#### **6.7.3.1** Progression free survival

Progression free survival may be performed on the Safety Analysis Set set according to statistical methods defined in section §5.6.1.

#### 6.7.3.2 Overall survival

Overall survival may be performed on the Safety Analysis Set set according to statistical methods defined in section §5.6.1.

### 6.7.4 Progression / Relapse

The following items will be described by cohort and overall:

- Patients who progressed/relapsed
- For each progression/relapse
  - o Treatment received for progression/relapse
  - Response after additional treatments

### 6.7.5 New anti-cancer therapy given prior to disease progression

New anti-cancer therapy given prior to disease progression for lymphoma will be described.

- Patients with at least one new anti-cancer therapy given prior to disease progression
- Type of treatment: Immunotherapy, Chemotherapy, Radio-immunotherapy, Transplant and Other treatment
- Listings will be displayed for each type of treatment


### 6.8 Extent of exposure

The extent of exposure to study treatment will be performed on the Safety Analysis Set according to statistical methods defined in the section §5.6.1. No statistical test will be performed.

#### **6.8.1** Cycles

- Duration of treatment
- Cycles performed
- Number of cycles performed

#### 6.8.2 Dose

The following items will be described:

- Cumulative total dose
  - Dose intensity
- Relative dose intensity

#### 6.8.3 Dose modifications

Dose delays, infusion interruptions, and drug withdrawals will be described by cycle and overall.

### 6.9 Safety analysis

Safety analysis will also be performed on the Safety Analysis Set according to statistical methods defined in the section §5.6.1. No statistical test will be performed.

#### **6.9.1** Treatment Emergent Adverse Events

Treatment emergent adverse event (TEAE) is defined as an AE that had an onset date or a worsening in severity from baseline (pre-treatment) on or after the first dose of study drug up to 90 days following study drug discontinuation, regardless of whether or not the patient starts a new anti-lymphoma therapy. TEAEs also include all irAEs and drug-related serious AEs recorded up to 90 days after the last dose of study drug. Treatment-related AEs include those events considered by the investigator to be definitely, possibly, or probably related to study treatment or with missing assessment of the causal relationship.

- Patients with at least one event:
  - TEAEs
  - TEAEs of grade ≥ 3
  - TEAEs leading to treatment discontinuation or interruption
  - Fatal TEAEs
  - irAE
- Number of TEAEs by patient, overall and by cohort
- Patients with at least one event and number of events by SOC and PT:
  - TEAEs: overall and by highest grade
  - o TEAEs of grade ≥ 3
  - TEAEs leading to treatment discontinuation or interruption: overall and by highest grade
  - Fatal TEAE (with listings)

- Patients with at least one treatment emergent AESI and number of events by type of special interest and PT (with listings)
- Patients with at least one irAE and number of events by type of irAE and PT:
  - with grade ≥ 3 (with listing)
  - o all grade (with listing), only for final analysis
- Characteristics of TEAEs overall and cohort: onset intensity, highest intensity, outcome, relationship to study drug, action taken with study drug

#### 6.9.2 Serious Adverse Events

- Patients with at least one event:
  - Serious TEAE
  - Serious TEAEs leading to treatment discontinuation or interruption
- Patients with at least one event and number of events by SOC and PT:
  - Serious TEAE: overall and by highest grade
  - Serious TEAEs leading to treatment discontinuation or interruption: overall and by highest grade
- Characteristics of serious TEAEs overall and cohort: onset intensity, highest intensity, outcome, relationship to study drug, action taken with study drug
- Listing of Serious TEAE

### 6.9.3 Secondary primary malignancies

The following items will be described:

- Patients with at least one other malignancy
- Other malignancies by SOC/PT
- Time to onset other malignancies from inclusion
- Narratives of other malignancies

### 6.9.4 Deaths

- Number of patients who died: overall and by period of death (before/during/after treatment)
- Cause of death and disease status by period of death
- Listing of patients who died
- Narratives of fatal SAEs

#### 6.9.5 Clinical Laboratory / Vital signs

Shift from baseline to worst baseline grade will be presented for clinical laboratories.

Summary of Increase in 2 or More CTCAE Toxicity Grades as Compared with Baseline

Vital sign (temperature, blood pressure, and pulse) will be presented for treatment period and safety follow-up.

Version 1.0 - 12APR2023

#### 6.9.6 Pregnancies

Narratives of pregnancies will be displayed by cohort.

### 6.10 Concomitant treatments

### 6.10.1 Prior treatment reported at enrollment

Prior treatments reported at enrollment will be described.

Prior treatments are defined as medications that stopped before the first dose of study drug.

#### **6.10.2** Concomitant treatments

Concomitant treatments during treatment period will be described.

- Patients with at least one concomitant treatment during treatment period
- Concomitant treatments received during treatment period will be listed

Concomitant treatments are defined as medications that

 started before the first dose of study drug and were continuing at the time of the first dose of study drug

or

- started on or after the date of the first dose of study drug up to 30 days after the patient's last dose.


## **7 STATISTICAL OUTPUTS**

All sections except subsections 7.1 Study sSummary, 7.4 Major protocol deviation Except mentionned otherwise, the header for all subsections will be as follows:

| Safety Analysis Set | | |
|---------------------|----------|-------|
| Cohort 1 | Cohort 2 | Total |
| N=XX | N=XX | N=XX |

### Subsection 7.1 Study summary and 7.4 Major protocol deviation

Except mentionned otherwise, the header will be as follows:

| Enrolled Set | | |
|--------------|----------|-------|
| Cohort 1 | Cohort 2 | Total |
| N=XX | N=XX | N=XX |

# 7.1 Study Summary

### 7.1.1 Overall description

Table 7.1-1 Number of patients by country and by center - Enrolled set

| | Header |
|--------------------|-------------|
| Number of patients | XXX (XX.X%) |
| Country | |
| XXXX | XXX (XX.X%) |
| XXXX | XXX (XX.X%) |
| XXXX | XXX (XX.X%) |
| Center name | |
| XXXX | XXX (XX.X%) |
| XXXX | XXX (XX.X%) |
| XXXX | XXX (XX.X%) |

Table 7.1-2 Number of patients at each timepoint - Safety Analysis set

| | Header |
|-----------------------------|-------------|
| Baseline | XXX (XX.X%) |
| During treatment | XXX (XX.X%) |
| End of treatment evaluation | XXX (XX.X%) |
| Safety follow-up | XXX (XX.X%) |
| Efficacy follow-up | XXX (XX.X%) |

## 7.1.2 Study dates

Table 7.1-3 Inclusion dates - Enrolled sets

| | Header |
|------------------------|------------|
| Inclusion dates | |
| First inclusion | XX/XX/XXXX |
| Last inclusion | XX/XX/XXXX |
| Safety analysis set | |
| First cycle day 1 date | XX/XX/XXXX |
| Last cycle day 1 date | XX/XX/XXXX |

Table 7.1-4 Date of last visit last patient - Enrolled set

| | Header |
|-------------------------|------------|
| Last Visit Last Patient | XX/XX/XXXX |

Last visit includes visits performed during follow-up period.

#### 7.1.3 Follow-up duration

Table 7.1-5 Follow-up duration - Safety Analysis set

| table 7.1-3 Follow-up duration - Safety Analysis set | | | | | | | |
|---|---|---|---|---|---|---|---|
| | Cohort | N | Median | 95% Confidence Limits | | Min | Max |
| | | | | Lower | Upper | | |
| Follow-up duration | Cohort 1 | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| (months) | Cohort 2 | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Total Safety | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Analysis Set | | | | | | |

Follow-up duration is based on OS since inclusion until last contact date and calculated with a reverse Kaplan Meier method.

# 7.2 Study patients

# 7.2.1 Disposition of patients

Table 7.2-1 Permanent treatment discontinuation during the study - Safety Analysis set

| | Header |
|--------------------------------------------------------|--------------|
| Permanent treatment discontinuation | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, reason for permanent treatment discontinuation | |
| Progressive disease | XX (XX.X%) |
| Adverse event | XX (XX.X%) |
| Death | XX (XX.X%) |
| Withdrawal by subject | XX (XX.X%) |
| Protocol violation | XX (XX.X%) |
| Physician decision | XX (XX.X%) |
| Other | XX (XX.X%) |
| If yes, last cycle performed | |
| Cycle 1 | XX (XX.X%) |
| | XX (XX.X%) |
| Time between inclusion and withdrawal (months) | |
| Number | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | xx;xx |

Figure 1: Disposition of patients



Listing 7.2-1 Permanent treatment discontinuation - Safety Analysis Set (XX patients)

| Eisting 7.2 11 Climanent treatment discontinuation | | | | | | thene treatment discontinuation. Surety rimarysis set (1212 patients) | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Cohort | Patient | Sex | Age | Inclusion date | Number of | Permanent tr | Permanent treatment dis | |
| | | Identification<br>Number | | (years) | | cycles<br>received | Date | Reason | Specification |
| | X | XXX | X | XX | XX/XX/XXXX | X | XX/XX/XXXX | XXXX | XX |

Table 7.2-2 Patient status - Safety Analysis Set

| | Header |
|-----------------------------------------------|------------|
| Patient status | |
| Treatment ongoing | XX (XX.X%) |
| Efficacy follow-up | XX (XX.X%) |
| End of study | XX (XX.X%) |
| If end of study, reason | |
| Lost to Follow-Up | XX (XX.X%) |
| Withdrawal by subject | XX (XX.X%) |
| Death | XX (XX.X%) |
| Study termination | XX (XX.X%) |
| Physician decision | XX (XX.X%) |
| Major protocol violation | XX (XX.X%) |
| Other | XX (XX.X%) |
| If Other, Description of patient status other | |
| | XX (XX.X%) |

TIRHOL - Statistical Analysis Plan


# 7.2.2 Analysis Sets

Table 7.2-3 Patients included in the trial - Enrolled Set

| THE THE THE THE THE THE THE | tritti Emilia Set |
|-----------------------------|-------------------|
| | Header |
| Enrolled set | XX (XX.X%) |
| Safety Analysis Set | XX (XX.X%) |

<u>Listing 7.2-2 Patients excluded from Safety Analysis Set (XX patients)</u>

| Cohort | Cohort Patient identification Safety A | | Patient identification Safety Analysis Inclusion Received at least one | | | Received at least one | Informed consent | Date of signature of |
|---|---|---|---|---|---|---|---|---|
| | number | Set | date | dose of Tislelizumab | | consent | | |
| X | X | No | | No | XXX | XX/XX/XXXX | | |

Figure 2: Analysis Sets



# 7.2.3 Analysis subsets

If applicable:

Table 7.2-4 Patients included in the trial with central confirmation of cHL diagnosis - Enrolled Set

| | Header |
|-------------------|------------|
| Confirmed cHL set | XX (XX.X%) |

<u>Listing 7.2-3 Patients excluded from Confirmed cHL Set (XX patients)</u>

| Cohort | Patient identification | Safety Analysis | Confirmed Set | Inclusion | Informed | Date of signature of | Local | Central |
|---|---|---|---|---|---|---|---|---|
| | number | Set | | date | consent | consent | diagnosis | diagnosis |
| X | X | X | No | | XXX | XX/XX/XXXX | | |

# 7.3 Inclusion / Exclusion criteria

#### Inclusion criteria:

Patients may be enrolled in the study only if they meet all of the following criteria:

- 1. Male or female ≥ 18 years of age at time of informed consent (or acceptable age according to local regulations, whichever is older)
- 2. Histologically confirmed diagnosis of relapsed or refractory cHL
- 3. Relapsed cHL (disease progression after PR or CR to the most recent therapy) or refractory cHL (failure to achieve PR or CR to most recent therapy). Patients will be allocated to one of two cohorts based on the following criteria:
  - Cohort 1: Relapsed or refractory to prior autologous hematopoietic stem cell transplant (HSCT)
    - Has failed to achieve a response or has had disease progression after autologous HSCT
    - Is not a candidate for additional autologous or allogeneic HSCT
  - Cohort 2: Relapsed or refractory to salvage chemotherapy and has not received prior autologous or allogeneic HSCT
    - Has received at least 1 prior systemic regimen for cHL
    - Is not a candidate for autologous or allogeneic HSCT
- 4. Measurable disease defined as  $\geq$  1 FDG-avid nodal lesion that is > 1.5 cm in the longest diameter, or  $\geq$  1 FDG-avid extra-nodal lesion (eg, hepatic nodules) that is > 1 cm in the longest diameter
- 5. Able to provide fresh or archival tumor tissues (formalin-fixed paraffin-embedded [FFPE] blocks or approximately 15 freshly cut, unstained FFPE slides) from an evaluable core or excisional biopsy with an associated pathological report
- 6. ECOG performance status of 0 or 1
- 7. Life expectancy ≥ 12 weeks
- 8. Adequate organ function, as indicated by the following laboratory values:
  - a. Absolute neutrophil count (ANC)  $\geq$  1.0 x 109/L, independent of growth factor support within 7 days of first dose
  - b. Platelet ≥ 75 x 109/L, independent of growth factor support within 7 days of first dose
  - c. Hemoglobin (Hgb) ≥ 8 g/dL or ≥ 5 mmol/L
  - d. Creatinine clearance > 30 mL/min
  - e. AST (SGOT) and ALT (SGPT)  $\leq$  2.5 x the ULN or  $\leq$  5 x ULN if liver lymphoma involvement is present
  - f. Serum total bilirubin  $\leq$  1.5 x ULN (total bilirubin level < 4 x ULN for patients with Gilbert syndrome)
- 9. No evidence of dyspnea at rest and a pulse oximetry of > 92% while breathing room air
- DLCO (adjusted for alveolar volume) > 60% of predicted value; FEV1 and FVC, FEV1/ FVC all > 50% predicted value
- 11. Female patients of childbearing potential must be willing to use a highly effective method of contraception for the duration of the study and for ≥ 120 days after the last dose of tislelizumab, and have a negative urine or serum pregnancy test within 7 days before the first dose of study drug.
- 12. Males are eligible to enter and participate in the study if they have been vasectomized or if they agree to use barrier contraception with other highly effective methods during the study treatment period and for ≥ 120 days after the last dose of tislelizumab
- 13. Ability to provide written informed consent and can understand and comply with the requirements of the study


#### Exclusion criteria:

Patients will not be enrolled in the study if they meet any of the following criteria:

- 1. Nodular lymphocyte-predominant Hodgkin lymphoma or gray zone lymphoma
- 2. Prior allogeneic hematopoietic stem cell transplantation
- 3. History of severe hypersensitivity reaction to monoclonal antibodies
- 4. New York Heart Association (NYHA) class III or IV heart failure, unstable angina, severe uncontrolled ventricular arrhythmia, electrocardiographic evidence of acute ischemia, or myocardial infarction within 6 months of first day of screening
- 5. Prior malignancy within the past 3 years except for curatively treated basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast, or other site for which in situ carcinoma has metastatic potential
- 6. Prior therapy targeting PD-1 or PD-L1, anti-PD-L2, or anti CTLA-4 pathways
- 7. Has received:
  - Systemic chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to Cycle 1 Day 1
  - Recent treatment with another monoclonal antibody within 4 weeks prior to Cycle 1 Day 1
  - Investigational treatment or device within 4 weeks (or 5 half-lives, whichever is shorter) prior to Cycle 1 Day 1
  - Or has not recovered from AEs (ie, ≤ Grade 1 or baseline level) due to prior therapy. (Note: Patients with alopecia or ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study if all other criteria are met)
- 8. Active autoimmune disease or history of autoimmune disease that may relapse
  - Patients with the following are not excluded and may proceed to further screening: Vitiligo, eczema, type I diabetes mellitus, and endocrine deficiencies including thyroiditis managed with replacement hormone and/or physiologic corticosteroids
  - Patients with the following should be evaluated for the presence of target organ involvement and the potential need for systemic treatment, but should otherwise be eligible: Rheumatoid arthritis and/or other arthropathies, Sjögren's syndrome, or psoriasis controlled with topical medication, and patients with positive serology such as positive antinuclear antibody or antithyroid antibody
- 9. Conditions requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of the first dose of tislelizumab Note: Patients with the following are not excluded and may proceed to further screening:
  - Adrenal replacement doses of ≤ 10 mg daily prednisone equivalent in the absence of active autoimmune disease
  - Topical, ocular, intra-articular, intranasal, and inhalational corticosteroid (with minimal systemic absorption)
  - A brief course of corticosteroid for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen)
- 10. History of interstitial lung disease or noninfectious pneumonitis or has evidence of interstitial lung disease or noninfectious pneumonitis
- 11. Serious acute or chronic infection requiring systemic therapy
- 12. Known central nervous system (CNS) lymphoma
- 13. Underlying medical conditions that, in the investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of toxicity or AEs
- 14. Known history of infection with HIV, human T-cell lymphotropic virus-1, or human T-cell lymphotropic virus-2
- 15. Serologic status reflecting active hepatitis B or C infection as follows:

- Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Patients with presence of HBcAb, but absence of HBsAg, are eligible only if hepatitis B virus (HBV) DNA is undetectable by an assay with sensitivity ≤ 20 IU/mL. If so, patients may either undergo regularly scheduled monitoring of HBV DNA or less frequent monitoring of HBV DNA while on prophylactic antiviral medication as defined by regional standard of care.
- Presence of hepatitis C virus (HCV) antibody. Patients with presence of HCV antibody are eligible only if HCV RNA is undetectable.
- 16. Autologous hematopoietic stem cell transplantation within 100 days of first dose of tislelizumab
- 17. CAR-T therapy within 12 months prior to the first dose of study drug
- 18. Use of any live vaccine against infectious diseases (eg, influenza, varicella, etc) within 4 weeks (28 days) of the first dose of tislelizumab, and any intended use within 60 days after the last dose of tislelizumab
- 19. Major surgery within 4 weeks of the first dose of tislelizumab
- 20. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
- 21. Has hypersensitivity to tislelizumab or any of its excipients
- 22. Concurrent participation in another therapeutic clinical trial

Table 7.3-1 Patients with at least one inclusion/exclusion criterion not fulfilled

| | Header |
|----------------------------------------------------|------------|
| Patients with at least one criterion not fulfilled | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Criterion not fullfilled | , , , |
| Inclusion criterion 01 | XX (XX.X%) |
| Inclusion criterion 02 | XX (XX.X%) |
| Inclusion criterion 03 | XX (XX.X%) |
| Inclusion criterion 04 | XX (XX.X%) |
| Inclusion criterion 05 | XX (XX.X%) |
| Inclusion criterion 06 | XX (XX.X%) |
| Inclusion criterion 07 | XX (XX.X%) |
| Inclusion criterion 08 | XX (XX.X%) |
| Inclusion criterion 09 | XX (XX.X%) |
| Inclusion criterion 10 | XX (XX.X%) |
| Inclusion criterion 11 | XX (XX.X%) |
| Inclusion criterion 12 | XX (XX.X%) |
| Inclusion criterion 13 | XX (XX.X%) |
| Exclusion criterion 01 | XX (XX.X%) |
| Exclusion criterion 02 | XX (XX.X%) |
| Exclusion criterion 03 | XX (XX.X%) |
| Exclusion criterion 04 | XX (XX.X%) |
| Exclusion criterion 05 | XX (XX.X%) |
| Exclusion criterion 06 | XX (XX.X%) |
| Exclusion criterion 07 | XX (XX.X%) |
| Exclusion criterion 08 | XX (XX.X%) |
| Exclusion criterion 09 | XX (XX.X%) |
| Exclusion criterion 10 | XX (XX.X%) |
| Exclusion criterion 11 | XX (XX.X%) |
| Exclusion criterion 12 | XX (XX.X%) |
| Exclusion criterion 13 | XX (XX.X%) |
| Exclusion criterion 14 | XX (XX.X%) |
| Exclusion criterion 15 | XX (XX.X%) |
| Exclusion criterion 16 | XX (XX.X%) |
| Exclusion criterion 17 | XX (XX.X%) |
| Exclusion criterion 18 | XX (XX.X%) |
| Exclusion criterion 19 | XX (XX.X%) |
| Exclusion criterion 20 | XX (XX.X%) |
| Exclusion criterion 21 | XX (XX.X%) |
| Exclusion criterion 22 | XX (XX.X%) |

Listing 7.3-1 Patients with at least one eligibility criterion not fulfilled - Safety Analysis Set (XX patients)

| Cohort | Patient identification number | Age (years) | Sex | Crite | <u>eria not fulfille</u> | d |
|---|---|---|---|---|---|---|
| | | | | Number | Description | Value |
| X | XXX | XXX | XX | XX | XXXXXX | XX |

# 7.4 Major protocol deviations

Table 7.4-1 Major protocol deviations - Enrolled set

| Table 7.4-1 Major proc | ocor ac mano |
|-------------------------------------------|--------------|
| | header |
| Patients with at least one major protocol | XX |
| deviation | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, type of major | |
| protocol deviation | |
| XXX | XX (XX.X%) |
| XXX | XX (XX.X%) |

<u>Listing 7.4-1 Patients with at least one major protocol deviation – Enrolled Set (XX patients)</u>

| Cohort* | Patient<br>identification<br>number | Inclusion date | Major<br>protocol<br>deviation | Safety<br>Analysis Set |
|---|---|---|---|---|
| X | XXXXX | XX/XX/XXXX | XXXX | XX |

# 7.5 Demographic and other baseline characteristics

# 7.5.1 Demographic characteristics

Table 7.5-1 Demographic characteristics at inclusion

| | Header |
|------------------------|--------------|
| Age (years) | |
| N | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Age group (years) | |
| <45 | XX (XX.X%) |
| >=45 | XX (XX.X%) |
| Sex | |
| Male | XX (XX.X%) |
| Female | XX (XX.X%) |
| Weight (kg) | |
| N | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Height (cm) | |
| N | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Body Surface Area (m²) | |
| N | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |

#### 7.5.2 Disease characteristics

#### 7.5.2.1 Diagnosis at inclusion

Table 7.5-2 Histological diagnosis according to local review

| 1 able 7.5-2 Histological diagnosis according | |
|-----------------------------------------------|--------------|
| | Header |
| Time since initial diagnosis (months) | |
| N | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |
| Initial histological diagnosis | |
| Classical Hodgkin Lymphoma | XX (XX.X%) |
| Other | XX (XX.X%) |
| Missing | XX |
| If Classical Hodgkin Lymphoma, subtype | |
| Nodular Sclerosis | XX (XX.X%) |
| Mixed Cellularity | XX (XX.X%) |
| Lymphocyte-depleted | XX (XX.X%) |
| Lymphocyte-rich | XX (XX.X%) |
| Unclassifiable | XX (XX.X%) |
| Missing | XX |
| If Other, specification | |
| XX | XX (XX.X%) |
| XX | XX (XX.X%) |
| Histological diagnosis at enrollment (local) | |
| Classical Hodgkin Lymphoma | XX (XX.X%) |
| Other | XX (XX.X%) |
| Missing | XX |
| If Classical Hodgkin Lymphoma, subtype | |
| Nodular Sclerosis | XX (XX.X%) |
| Mixed Cellularity | XX (XX.X%) |
| Lymphocyte-depleted | XX (XX.X%) |
| Lymphocyte-rich | XX (XX.X%) |
| Unclassifiable | XX (XX.X%) |
| Missing | XX |
| If Other, specification | |
| XX | XX (XX.X%) |
| XX | XX (XX.X%) |

Table 7.5-3 Histological diagnosis according to central review

| | Header |
|----------------------------------------------------|------------|
| Histological diagnosis according to central review | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If Yes, diagnosis | , , |
| XXX | XX (XX.X%) |
| XXX | XX (XX.X%) |

#### 7.5.2.2 Disease assessment at inclusion

Table 7.5-4 Disease assessments and staging at inclusion

| Table 7.5-4 Disease assessments and staging at inclusion | Header |
|----------------------------------------------------------|--------------|
| Patient status at time of enrollment | |
| Refractory | XX (XX.X%) |
| Relapse/Progressive | XX (XX.X%) |
| Ann Arbor stage | ` |
| I | XX (XX.X%) |
| II | XX (XX.X%) |
| III | XX (XX.X%) |
| IV | XX (XX.X%) |
| Unknown | XX (XX.X%) |
| Missing | XX |
| Performance Status (ECOG) | |
| Normal activities | XX (XX.X%) |
| Ambulatory able to carry out work | XX (XX.X%) |
| Ambulatory unable to carry out work | XX (XX.X%) |
| Confined to chair more than 50% of waking hours | XX (XX.X%) |
| Totally confined to chair | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Missing | XX |
| B symptoms | 777 |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Missing | XX |
| International Prognostic Score (Hasenclever) | 1.00 |
| 0 | XX (XX.X%) |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| 4 | XX (XX.X%) |
| 5 | XX (XX.X%) |
| 6 | XX (XX.X%) |
| 7 | XX (XX.X%) |
| Missing | XX (XX.X70) |
| International Prognostic Score (Hasenclever) in class | |
| 0-2 | XX (XX.X%) |
| >= 3 | XX (XX.X%) |
| Missing | XX |
| Bulky disease* | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Missing | XX (XX.X 70) |
| Erythrocyte Sedimentation Rate (ESR) (mm/hr) | 7// |
| N | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X (XX.XX) |
| Q1;Q3 | XX;XX |
| Min; Max | XX;XX |
| Till / Tim | /// / /// |

<sup>\*</sup>mediastinum/thorax ratio of 0.33 or size of any single node/nodal mass ≥ 10 cm in diameter

# 7.5.2.3 Prior therapy for cHL

Table 7.5-5 Number of prior lines of therapy for cHL

| | Header |
|------------------------------------------|--------------|
| Number of prior lines of therapy for cHL | |
| 1 | XX (XX.X%) |
| | XX (XX.X%) |
| Number of prior lines of therapy for cHL | |
| N | XX |
| Missing | |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Monoclonal antibody | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Missing | XX |
| Other immunotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Missing | XX |
| Chemotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Missing | XX |
| Radiotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Missing | XX |
| Autologous transplant | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Missing | XX |
| Other anti-cancer therapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Missing | XX |

#### 7.5.2.4 Nodal / Extra-nodal involvement at baseline

Table 7.5-6 Overview of nodal/extra-nodal involvement at baseline

| Table 7.5-6 Overview of house extra-nodar involvement at baseline | |
|---|---|
| | Header |
| Patients with at least one nodal involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Patients with at least one extra-nodal involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

EN-SOP-ST-03-Temp-01-SAP Template (Phase II/III) - V2.0 - Effective date: 14/12/2016

Table 7.5-7 Supra-diaphragmatic nodal involvement at baseline

| <u> Table 7.5-7 Supra-diaphragmatic nodal involve</u> | |
|-------------------------------------------------------|------------|
| | Header |
| Cervical right | i |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Cervical left | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Supraclavicular right | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Supraclavicular left | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Axillary right | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Axillary left | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Mediastinal | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |

Table 7.5-8 Infra-diaphragmatic nodal involvement at baseline

| | Header |
|-----------------|------------|
| Retroperitoneal | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Mesenteric | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Iliac right | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Iliac left | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Inguinal right | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Inguinal left | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |

Table 7.5-9 Other nodal involvement at baseline

| | Header |
|-------------------------|------------|
| Other nodal involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |

## <u>Listing 7.5-1 Patients with other nodal involvement localizations at baseline – Safety Analysis Set (XX</u>

patients)

| Cohort | Patient identification number | Other nodal involvement | Other nodal involvement -<br>localization |
|---|---|---|---|
| | | Yes | |

# Table 7.5-10 Extra-nodal involvement in the Head and Neck Area at baseline

| | Header |
|---------------|------------|
| Tonsil | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Cavum | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Parotid | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Orbit | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Sinus | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |

# Table 7.5-11 Extra-nodal involvement in Central Nervous System Area at baseline

| | Header |
|---------------|------------|
| Meningeal | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Other CNS | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |

Table 7.5-12 Extra-nodal involvement in the Digestive Tract Area at baseline

| | Header |
|----------------------|------------|
| Stomach | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Duodenum | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Small Intestine | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Ileo-caecal junction | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Colon | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Rectum | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |

| | Header |
|-------------------------------|--------------------------|
| Liver | |
| Li <b>ver</b><br>Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| | ^^ (^^.^ <sup>70</sup> ) |
| Pancreas<br>Normal | XX (XX.X%) |
| Involved<br>Not Evaluated | XX (XX.X%) |
| | XX (XX.X%) |
| Pleura | VOV (VOV VOV ) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Lung | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Ascites | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Pericardium | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Breast | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Gonadal | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Kidney | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Adrenal | (/3/////0) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Thyroid | ^^ (^^.^*0) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%)<br>XX (XX.X%) |
| Not Evaluated | XX (XX.X%)<br>XX (XX.X%) |
| | AA (AA.A%) |
| Skin<br>Normal | VV (VV V0/) |
| | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Soft Tissues | 101 /101 101 |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Bone | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Blood | , |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Other extra-nodal involvement | 121 (1211/10) |
| No | XX (XX.X%) |

TIRHOL - Statistical Analysis Plan


# <u>Listing 7.5-2 Patients with other extra-nodal involvement localizations at baseline – Safety Analysis Set</u>

(XX patients)

| Coh | ort* | Patient<br>identification<br>number | Other extra-nodal involvement | Other extra-nodal involvement -<br>localization |
|---|---|---|---|---|
| | | | Yes | |

#### 7.5.3 Tumor assessment

# 7.5.3.1 PET scan at baseline

Table 7.5-14 PET scan at baseline

| | Header |
|---------------------------------------------|-------------|
| PET scan performed at baseline | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, bone marrow involved : | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, presence of hypermetabolic lesion : | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| If yes, SUVmax : | |
| N | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |

#### 7.5.3.2 CT scan at baseline

Table 7.5-15 Sites and methods used for tumor assessment at baseline

| | Header |
|----------------------------------|-------------|
| Tumor assessment | |
| CT scan performed at baseline | |
| Not Done | XX (XX.X%) |
| Done | XX (XX.X%) |
| If yes, number of sites used for | |
| esponse evaluation | |
| Ň | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |

SPD: Sum of the Product of the Diameters

Table 7.5-16 Methods of measurements at baseline

| | Header |
|-------------------------------------|------------|
| Methods of measurements at baseline | |
| Clinical Examination | XX (XX.X%) |
| CT Scan | XX (XX.X%) |
| Ultrasound | XX (XX.X%) |
| NMR/MRT/MRI | XX (XX.X%) |
| CT/PET Scan | XX (XX.X%) |
| Other | XX (XX.X%) |

N : Number of sites

Table 7.5-17 Extra-nodal sites evaluable but not measurable at baseline

| | Header |
|-------------------------------------------------------|--------------|
| Patients with at least one extra-nodal site evaluable | |
| but not measurable | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Number of extra-nodal sites evaluable but | |
| not measurable per patient | |
| N | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min; Max | XX;XX |

# 7.5.4 Medical history

#### Table 7.5-18 Medical history

| | Header |
|---|---|
| At least one medical history | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, category* | |
| Prior cancer history | XX (XX.X%) |
| Other relevant medical history | XX (XX.X%) |
| If other prior cancer, at least one persisting other cancer history | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If other medical history, at least one persisting other relevant medical history | ' ' |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

<sup>\*</sup> The sum of category can be > 100% because categories are not mutually exclusive

# Table 7.5-19 Relevant medical history (including prior cancer) by SOC/PT

| System | Organ | Class | H | leader |
|---|---|---|---|---|
| Preferred Term | 1 | | | |
| Patients with a le | east one relevant medical history | | XX | (XX.X%) |
| SOC1 | | | XX | (XX.X%) |
| PT1 | | | XX | (XX.X%) |
| PT2 | | | XX | (XX.X%) |
| | | | XX | (XX.X%) |
| SOC2 | | | XX | (XX.X%) |
| PT1 | | | XX | (XX.X%) |
| PT2 | | | XX | (XX.X%) |
| | | | XX | (XX.X%) |

# Listing 7.5-3 Relevant medical history (including prior cancer) - Safety Analysis Set (XX patients)

| Cohort | Patient identification number | Inclusion date | Category | Type of prior cancer/disease | Disease onset date | Persisting | Grade | End date |
|---|---|---|---|---|---|---|---|---|
| X | XX | XX/XX/XXXX | XX | XX | XX/XX/XXXX | XX | XX | XX/XX/XXXX |

# 7.5.5 Vital signs

Table 7.5-20 Vital signs at baseline

| <u> Fable 7.5-20 Vital signs at baseline</u> | |
|----------------------------------------------|-------------|
| | Header |
| Vital sign examination performed | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Systolic blood pressure (mmHG) | |
| N | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Diastolic blood pressure (mmHG) | |
| N | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Pulse (beats/min) | |
| N | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Body temperature (°C) | |
| N | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |

#### 7.5.6 Other clinical exams

Table 7.5-21 Clinical examination at baseline

| | Header |
|----------------------------------|------------|
| Clinical examination | |
| Not done | XX (XX.X%) |
| Done | XX (XX.X%) |
| If done, result | |
| Abnormal | XX (XX.X%) |
| Normal | XX (XX.X%) |
| If abnormal, due to active lymph | oma |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If abnormal, due to study treatn | nent |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If abnormal, due to other reason | 1 |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

<u>Listing 7.5-4 Patients with abnormal clinial exam at baseline - Safety Analysis Set (XX patients)</u>

| Cohort | Patient | Inclusion | | Clinical exam | |
|---|---|---|---|---|---|
| | identification<br>number | date | Date | Result | Specify reason |
| | | | | Abnormal | |

| <u> Fable 7.5-22 Serologies at baseline</u> | |
|---------------------------------------------|------------|
| | Header |
| HIV Serology | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not done / Missing | XX |
| HCV Serology | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not done / Missing | XX |
| HBV serology | |
| HBs Ag | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not done / Missing | XX |
| Anti HBs | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not done / Missing | XX |
| Anti HBc | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not done / Missing | XX |
| Vaccination | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Unknown | XX |

Table 7.5-23 Cardiac exam at baseline

| | Header |
|----------------------------------------|-------------|
| Electrocardiogram | |
| Not done | XX (XX.X%) |
| Done | XX (XX.X%) |
| If done, result | |
| Normal | XX (XX.X%) |
| Clinically significant abnormality | XX (XX.X%) |
| Non clinically significant abnormality | XX (XX.X%) |
| Echocardiography / Isotopic method | |
| Not done | XX (XX.X%) |
| Done | XX (XX.X%) |
| If done, result | ' ' |
| Normal | XX (XX.X%) |
| Abnormal | XX (XX.X%) |
| If done, LVEF (%) | , , |
| N | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Cardiac biomarkers | |
| Not done | |
| Done | |
| If done, Troponin I | |
| Normal | XX (XX.X%) |
| Above limit | XX (XX.X%) |
| If done, Troponin T | |
| Normal | XX (XX.X%) |
| Above limit | XX (XX.X%) |

Listing 7.5-5 Patients with abnormal cardiac exam at baseline - Safety Analysis Set (XX patients)

| Cohort | Patient | Inclusion | Echocardiography / Isotopic method | | |
|---|---|---|---|---|---|
| | identification<br>number | date | Date | Result | If abnormal,<br>specify |

**Table 7.5-24 Childbearing potential** 

| | Header |
|----------------------------------|------------|
| Female of childbearing potential | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, pregnancy test | |
| Done | XX (XX.X%) |
| Not done | XX (XX.X%) |
| If done, result | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |

Table 7.5-25 Pulmonary function test

| Header |
|---|
| No XX (XX.X%) Yes XX (XX.X%) If yes, FEV1 (L) XX N XX Mean (SD) XX.X (XX.X) Median XX.X |
| No XX (XX.X%) Yes XX (XX.X%) If yes, FEV1 (L) XX N XX Mean (SD) XX.X (XX.X) Median XX.X |
| If yes, FEV1 (L) N Mean (SD) Median XX XX.X (XX.X) XX.X (XX.X) |
| N XX Mean (SD) XX.X (XX.X) Median XX.X |
| N XX Mean (SD) XX.X (XX.X) Median XX.X |
| Median XX.X |
| 01 - 03 |
| Q1; Q3 XX; XX |
| Min ; Max XX ; XX |
| If yes, FEV1 Best/Pred (%) |
| N XX |
| Mean (SD) XX.X (XX.X) |
| Median XX.X |
| Q1 ; Q3 XX ; XX |
| Min ; Max XX ; XX |
| If yes, FVC (L) |
| N XX |
| Mean (SD) XX.X (XX.X) |
| Median XX.X |
| Q1; Q3 XX; XX |
| Min; Max XX; XX |
| If yes, FVC Best/Pred (%) |
| N XX |
| Mean (SD) XX.X (XX.X) |
| Median XX.X |
| Q1; Q3 XX; XX |
| Min; Max XX; XX |
| If yes, DLCOc-SB Best/Pred (%) |
| N XX |
| Mean (SD) XX.X (XX.X) |
| Median XX.X |
| Q1;Q3 XX;XX |
| Min; Max XX; XX |
| If yes, FEV1/FVC (%) |
| N XX |
| Mean (SD) XX.X (XX.X) |
| Median XX.X |
| Q1; Q3 XX; XX |
| Min; Max XX; XX |
| If yes, pulse oximetry (%) |
| N XX |
| Mean (SD) XX.X (XX.X) |
| Median XX.X |
| Q1; Q3 XX; XX |
| Min; Max XX; XX |

# 7.6 Evaluation during study

#### 7.6.1 Clinical examination

7.6.1.1 During treatment

Table 7.6-1 Clinical examination by cycle during treatment

| Clinical Examination | Header |
|----------------------|------------|
| Cycle 1 | |
| Normal | XX (XX.X%) |
| Abnormal | XX (XX.X%) |
| Not done / Missing | XX |
| Cycle 2 | |
| Normal | XX (XX.X%) |
| Abnormal | XX (XX.X%) |
| Not done / Missing | `XX |
| ••• | |

<u>Listing 7.6-1 Patients with abnormal clinial exam due to active lymphoma during treatment - Safety</u>

Analysis Set (XX patients)

| - 1 | 22200 | TALL PROTECTION | _ | | | | |
|---|---|---|---|---|---|---|---|
| | Cohort | Patient | Age at | Inclusion | Clinical exam | | |
| | | identification<br>number | inclusion<br>(years) | date | Date | Result | Specify reason |
| | | | | | | Abnormal | |

Table 7.6-2 Performance status (ECOG) by cycle during treatment

| Performance<br>(ECOG) | Status | Header |
|-----------------------|--------|------------|
| Cycle 1 | | |
| 0 | | XX (XX.X%) |
| 1 | | XX (XX.X%) |
| 2 | | XX (XX.X%) |
| 3 | | XX (XX.X%) |
| Missing | | XX |
| Cycle 2 | | |
| 0 | | XX (XX.X%) |
| 1 | | XX (XX.X%) |
| 2 | | XX (XX.X%) |
| 3 | | XX (XX.X%) |
| 4 | | XX (XX.X%) |
| Missing | | XX |

#### 7.6.1.2 At end of treatment (safety follow-up)

Table 7.6-3 Clinical examination by cycle at end of treatment

| Clinical Examination | Header |
|----------------------------------------|------------|
| End of treatment –<br>Safety follow-up | |
| Normal | XX (XX.X%) |
| Abnormal | XX (XX.X%) |
| Not done / Missing | XX |


# <u>Listing 7.6-2 Patients with abnormal clinial exam due to active lymphoma at end of treatment - Safety</u>

Analysis Set (XX patients)

| Г | Cohort | Patient | Age at | Inclusion -<br>date | Clinical exam | | am |
|---|---|---|---|---|---|---|---|
| | | identification<br>number | inclusion<br>(years) | | Date | Result | Specify reason |
| | | | | | | Abnormal | |

Table 7.6-4 Performance status (ECOG) by cycle at end of treatment

| Performance Status<br>(ECOG) | Header |
|----------------------------------------|------------|
| End of treatment –<br>Safety follow-up | |
| 0 | XX (XX.X%) |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| Missing | XX |

#### 7.6.1.3 During Efficacy follow up

Table 7.6-5 Clinical examination by cycle during efficacy follow-up

| Clinical Examination | Header |
|----------------------|------------|
| EFFICACY FOLLOW-UP 1 | |
| Normal | XX (XX.X%) |
| Abnormal | XX (XX.X%) |
| Not done / Missing | XX |
| EFFICACY FOLLOW-UP 2 | |
| Normal | XX (XX.X%) |
| Abnormal | XX (XX.X%) |
| Not done / Missing | XX |

Listing 7.6-3 Patients with abnormal clinial exam due to active lymphoma during efficacy follow-up -

Safety Analysis Set (XX patients)

| Cohort | Patient | Age at | Inclusion | Clinical exam | | m |
|---|---|---|---|---|---|---|
| | identification<br>number | inclusion<br>(years) | date | Date | Result | Specify reason |
| | | | | | Abnormal | |

Table 7.6-6 Performance status (ECOG) by cycle during efficacy follow-up

| Performance Status | Header |
|--------------------|------------|
| (ECOG) | |
| Visit 1 | |
| 0 | XX (XX.X%) |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| Missing | XX |
| Visit 2 | |
| 0 | XX (XX.X%) |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| Missing | XX |

# 7.6.2 Tumor assessment

7.6.2.1 During treatment and efficacy follow-up

Table 7.6-7 PET scan at each visit during treatment

| | Header |
|-------------------------------|----------------------------------------|
| DET | |
| PET scan | |
| PET scan done at evaluation 1 | \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, bone marrow involved | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Deauville criteria | |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| 4 | XX (XX.X%) |
| 5 | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| If yes, localization of most | |
| hypermetabolic lesion : | |
| | XX (XX.X%) |
| SUVmax of most | |
| hypermetabolic lesion : | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1 ; Q3 | XX;XX |
| Min; Max | XX;XX |

Table 7.6-8 Sites and methods used for tumor assessment treatment

| | Header |
|----------------------------------|-------------|
| Tumor assessment | |
| Evaluation 1 | |
| Not Done | XX (XX.X%) |
| Done | XX (XX.X%) |
| If yes, number of sites used for | |
| response evaluation | |
| N N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| If yes, SPD difference from | |
| baseline (%) | |
| N N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| <b></b> | |

SPD: Sum of the Product of the Diameters

Table 7.6-9 Methods of measurements during treatment

| | Header |
|-----------------------------------------|------------|
| Methods of measurements at evaluation 1 | |
| Clinical Examination | XX (XX.X%) |
| CT Scan | XX (XX.X%) |
| Ultrasound | XX (XX.X%) |
| NMR/MRT/MRI | XX (XX.X%) |
| CT/PET Scan | XX (XX.X%) |
| Other | XX (XX.X%) |

N : Number of sites

Table 7.6-10 Extra-nodal sites evaluable but not measurable during treatment

| Patients with at least one extra-nodal site evaluable but not measurable | Header |
|---|---|
| At evaluation 1 | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Number of extra-nodal sites | |
| evaluable but not measurable per patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |

Table 7.6-11 Significant increase in size of non target lesion(s) during treatment

| Significant increase in size of non target lesion(s) | Header |
|------------------------------------------------------|--------------|
| Significant increase in size of non target | |
| lesion(s) at evaluation 1 | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, number of significant increase in | |
| size of non target lesion(s) per patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |

Table 7.6-12 New lymphoma lesion(s) during treatment

| | Header |
|------------------------------------------|--------------|
| New lymphoma lesion(s) | |
| New lymphoma lesion(s) from screening at | |
| evaluation 1 | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Number of new lymphoma | |
| lesion(s) per patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |

Table 7.6-13 Spleen and liver assessment during treatment

| | Header |
|----------------------------|------------|
| Evaluation at evaluation 1 | |
| Not done | XX (XX.X%) |
| Done | XX (XX.X%) |
| If yes, spleen enlarged | |
| Yes | XX |
| No | XX |
| If yes, liver enlarged | |
| Yes | XX |
| No | XX |

Table 7.6-14 Methods of spleen and liver assessment during treatment

| | Header |
|-----------------------------------------|------------|
| Methods of measurements at evaluation 1 | |
| Clinical Examination | XX (XX.X%) |
| CT Scan | XX (XX.X%) |
| Ultrasound | XX (XX.X%) |
| NMR/MRT/MRI | XX (XX.X%) |
| CT/PET Scan | XX (XX.X%) |
| Other | XX (XX.X%) |
| If other, specification | |
| | XX (XX.X%) |

Table 7.6-15 Metabolic response during treatment

| | Header |
|-----------------------------------------------------------|------------|
| Metabolic response (PET -CT-based) | |
| Metabolic response according to Lugano | |
| classification (PET-CT-scan) at evaluation 1 | |
| Complete metabolic response | XX (XX.X%) |
| Partial metabolic response | XX (XX.X%) |
| No metabolic response | XX (XX.X%) |
| Progressive metabolic disease | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| If progressive metabolic disease, Response | |
| according to LYRIC classification (PET-CT-based) | |
| Complete response | XX (XX.X%) |
| Partial response | XX (XX.X%) |
| Stable disease | XX (XX.X%) |
| Progressive disease | XX (XX.X%) |
| Indeterminate response | XX (XX.X%) |
| Not evaluable | XX (XX.X%) |
| If indeterminate response | |
| IR1 - >=50% increase in SPD in first 12 weeks | XX (XX.X%) |
| IR2 - <50% increase in SPD with new lesion or ≥50% | XX (XX.X%) |
| increase in PPD of a lesion or set of lesions at any time | |
| during treatment | |
| IR3 - increase in FDG uptake without a concomitant | XX (XX.X%) |
| increase in lesion size meeting criteria for PD | |

Table 7.6-16 Radiologic response according to Lugano classification (CT-based) during treatment

| | Header |
|--------------------------------------------|------------|
| Radiologic according to Lugano (CT- | |
| based) | |
| Radiologic response at evaluation 1 | |
| Complete radiologic response | XX (XX.X%) |
| Partial remission | XX (XX.X%) |
| Stable disease | XX (XX.X%) |
| Progressive disease | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| If progressive radiologic disease, | |
| Response according to LYRIC | |
| classification (CT-based) | |
| Complete response | XX (XX.X%) |
| Partial response | XX (XX.X%) |
| Stable disease | XX (XX.X%) |
| Progressive disease | XX (XX.X%) |
| Indeterminate response | XX (XX.X%) |
| Not evaluable | XX (XX.X%) |
| If indeterminate response | , , |
| IR1 - >=50% increase in SPD in first 12 | XX (XX.X%) |
| weeks | , , |
| IR2 - <50% increase in SPD with new | XX (XX.X%) |
| lesion or ≥50% increase in PPD of a lesion | |
| or set of lesions at any time during | |
| treatment | |

# 7.6.2.2 At end of treatment (safety follow-up)

# Table 7.6-17 PET scan at each visit at end of treatment

| | Header |
|------------------------------|---------------|
| DET | |
| PET scan | |
| PET scan done at end of | |
| treatment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, bone marrow | |
| involved | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Deauville criteria | |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| 4 | XX (XX.X%) |
| 5 | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| If yes, localization of most | ` ′ |
| hypermetabolic lesion: | |
| | XX (XX.X%) |
| | 701 (7010177) |
| SUVmax of most | |
| hypermetabolic lesion: | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1;Q3 | XX ; XX |
| 2 , 2 | XX;XX |
| Min ; Max | ^^ , ^^ |

EN-SOP-ST-03-Temp-01-SAP Template (Phase II/III) - V2.0 - Effective date: 14/12/2016

Table 7.6-18 Sites and methods used for tumor assessment treatment at end of treatment

| | Header |
|----------------------------------|-------------|
| Tumor assessment | |
| Evaluation at end of treatment | |
| Not Done | XX (XX.X%) |
| Done | XX (XX.X%) |
| If yes, number of sites used for | |
| esponse evaluation | |
| Ň | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| If yes, SPD difference from | |
| baseline (%) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |

SPD: Sum of the Product of the Diameters

Table 7.6-19 Methods of measurements at end of treatment

| | Header |
|---------------------------------------------|------------|
| Methods of measurements at end of treatment | |
| Clinical Examination | XX (XX.X%) |
| CT Scan | XX (XX.X%) |
| Ultrasound | XX (XX.X%) |
| NMR/MRT/MRI | XX (XX.X%) |
| CT/PET Scan | XX (XX.X%) |
| Other | XX (XX.X%) |

N : Number of sites

Table 7.6-20 Extra-nodal sites evaluable but not measurable at end of treatment

| Patients with at least one extra-nodal site evaluable but not measurable | Header |
|---|---|
| Evaluation at end of treatment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Number of extra-nodal sites | |
| evaluable but not measurable per patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |

Table 7.6-21 Significant increase in size of non target lesion(s) at end of treatment

| Significant increase in size of non target | Header |
|---------------------------------------------|--------------|
| lesion(s) | |
| Significant increase in size of non target | |
| lesion(s) at end of treatment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Significant increase in size of non | |
| target lesion(s) per patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min; Max | XX;XX |

# Table 7.6-22 New lymphoma lesion(s) at end of treatment

| | Header |
|------------------------------------------|--------------|
| New lymphoma lesion(s) | |
| New lymphoma lesion(s) from screening at | |
| end of treatment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, New lymphoma lesion(s) per | |
| patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |

# Table 7.6-23 Spleen and liver assessment at end of treatment

| | Header |
|--------------------------------|------------|
| Evaluation at end of treatment | |
| Not done | XX (XX.X%) |
| Done | XX (XX.X%) |
| If yes, spleen enlarged | |
| Yes | XX |
| No | XX |
| If yes, liver enlarged | |
| Yes | XX |
| No | XX |

# Table 7.6-24 Methods of spleen and liver assessment at end of treatment

| | Header |
|---------------------------------------------|------------|
| Methods of measurements at end of treatment | |
| Clinical Examination | XX (XX.X%) |
| CT Scan | XX (XX.X%) |
| Ultrasound | XX (XX.X%) |
| NMR/MRT/MRI | XX (XX.X%) |
| CT/PET Scan | XX (XX.X%) |
| Other | XX (XX.X%) |
| If other, specification | |
| | XX (XX.X%) |

Table 7.6-25 Metabolic response at end of treatment

| <u>onse at en</u> |
|-------------------|
| Header |
| XX (XX.X%) |
| ' ' |

Table 7.6-26 Radiologic response according to Lugano classification (CT-based) at end of treatment

| | Header |
|-------------------------------------|------------|
| Radiologic according to Lugano | |
| (CT-based) | |
| Radiologic response at end of | |
| treatment | |
| Complete radiologic response | XX (XX.X%) |
| Partial remission | XX (XX.X%) |
| Stable disease | XX (XX.X%) |
| Progressive disease | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| If progressive radiologic | |
| disease, Response according | |
| to LYRIC classification (CT- | |
| based) | |
| Complete response | XX (XX.X%) |
| Partial response | XX (XX.X%) |
| Stable disease | XX (XX.X%) |
| Progressive disease | XX (XX.X%) |
| Indeterminate response | XX (XX.X%) |
| Not evaluable | XX (XX.X%) |
| If indeterminate response | |
| IR1 - >=50% increase in SPD in | XX (XX.X%) |
| first 12 weeks | |
| IR2 - <50% increase in SPD | XX (XX.X%) |
| with new lesion or ≥50% in | |
| crease in PPD of a lesion or set of | |
| lesions at any time during | |
| treatment | |

#### 7.6.2.3 During efficacy follow-up

Table 7.6-27 Disease status during efficacy follow-up

| | Header |
|------------------------------------|------------|
| EFFICACY FOLLOW-UP 1 | |
| Change of diseasestatus since last | |
| visit | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, specification of change | ' |
| Progression | XX (XX.X%) |
| Improvement | XX (XX.X%) |
| If improvement, specification | ' ' |
| Complete response | XX (XX.X%) |
| Partial response | XX (XX.X%) |

# 7.7 Efficacy Analysis

#### 7.7.1 Primary efficacy endpoint analyses

#### 7.7.1.1 Main analysis

Table 7.7-1 ORR\* evaluation – Safety Analysis Set

| | Safety set |
|---------------------------------------------------|-----------------|
| Best response according to Lugano classification* | i |
| Complete Response | XX (XX.X%) |
| Partial Remission | XX (XX.X%) |
| Stable Disease | XX (XX.X%) |
| Progressive Disease | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| ORR according to Lugano classification** | |
| Patients with ORR | XX (XX.X%) |
| IC 90% for ORR rate | [XX.X% - XX.X%] |
| IC 95% for ORR rate | [XX.X% - XX.X%] |
| Binomial test *** | |
| Z test value | XX |
| One-sided p-value | X.XX |

Response of patients with no post-baseline response assessment (due to any reason) will be considered Not evaluated and patients will be considered non-responders.

EN-SOP-ST-03-Temp-01-SAP Template (Phase II/III) - V2.0 - Effective date: 14/12/2016

<sup>\*</sup>Lugano classification: for each evaluation, metabolic response (PET-CT based) if available, radiologic response (CT-based) otherwise

<sup>\*\*</sup>ORR is defined as the proportion of patients who achieve a best response of CR or PR per the Lugano Classification (Cheson et al 2014) from the first dose of Tislelizumab until data cut or the start of a new anti-lymphoma therapy and determined by the investigator

<sup>\*\*\*</sup> For analyses of primary endpoint

Version 1.0 – 12APR2023

Listing 7.7-1 Patients with best response "Not Evaluated" according to Lugano classification – Safety Analysis Set (XX patients)

| Disting / t/ I | I teremes with | a best res | pomse 1 | ot E / mateu | | CCOI GIII | C to Dagano | CICOSIII | CHULOII | Suret I I I I I | 313 500 (1111 | Juit Lie | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort | | | | Confirmed<br>cHL | Permanent treatment discontinuation | | | | | Evaluation | | New anti-lymp | homa therapy |
| | Patient<br>identification<br>number | Inclusion<br>date | Number<br>of cycles<br>received | | Date | Reason | Specification | Periode | Date | Metabolic<br>response<br>according to<br>Lugano<br>Classification<br>(PET-CT based) | Radiologic<br>response<br>according to<br>Lugano<br>Classification<br>(CT based) | Date | Туре |
| X | XXX | XX/XX/XXX | XX | XXX | XX/XX/ | XXXX | XXXX | XXX | XX/XX/X | XXX | XXX | XX/XX/XXXX | XXXXXX |
| | | X | | | XXXX | | | | XXX | | | | |
| | | | | | | | | XXX | XX/XX/X | XXX | XXX | XX/XX/XXXX | XXX |
| | l . | | | | | ı | | 1 | XXX | | | l | |
### 7.7.1.2 Sensitivity analysis

Table 7.7-2 ORR\* evaluation – Confirmed cHL Set

| | ••• |
|---------------------------------------------------|-------------------|
| | Confirmed cHL set |
| Best response according to Lugano classification* | |
| Complete Response | XX (XX.X%) |
| Partial Remission | XX (XX.X%) |
| Stable Disease | XX (XX.X%) |
| Progressive Disease | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| ORR according to Lugano classification** | |
| Patients with ORR | XX (XX.X%) |
| IC 90% for ORR rate | [XX.X% - XX.X%] |
| IC 95% for ORR rate | [XX.X% - XX.X%] |

Response of patients with no post-baseline response assessment (due to any reason) will be considered Not evaluated and patients will be considered non-responders.

Listing 7.7-2 Patients with best response "Not Evaluated" according to Lugano classification – Confirmed cHL Set (XX patients)

| Cohort | | | | Confirmed<br>cHL | Permanent treatment discontinuation | | Evaluation | | | New anti-lymphoma therapy | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Patient<br>identification<br>number | Inclusion<br>date | Number<br>of cycles<br>received | | Date | Reason | Specification | Periode | Date | Metabolic<br>response<br>according to<br>Lugano<br>Classification<br>(PET-CT based) | Radiologic<br>response<br>according to<br>Lugano<br>Classification<br>(CT based) | Date | Туре |
| X | XXX | XX/XX/XXX<br>X | XX | XXX | XX/XX/<br>XXXX | XXXX | XXXX | XXX | XX/XX/X<br>XXX | XXX | XXX | XX/XX/XXXX | XXXXXX |
| | | | | | | | | XXX | XX/XX/X<br>XXX | XXX | XXX | XX/XX/XXXX | XXX |

<sup>\*</sup>Lugano classification: for each evaluation, metabolic response (PET-CT based) if available, radiologic response (CT-based) otherwise

<sup>\*\*</sup>ORR is defined as the proportion of patients who achieve a best response of CR or PR per the Lugano Classification (Cheson et al 2014) from the first dose of Tislelizumab until data cut or the start of a new anti-lymphoma therapy and determined by the investigator

#### 7.7.1.3 Subgroup analyses

Table 7.7-3 ORR\* evaluation — Safety Analysis Set

| | Safety Analysis Set | |
|---|---|---|
| | Cohort 1 | Cohort 2 |
| Best response according to Lugano classification* | | |
| Complete Response | XX (XX.X%) | XX (XX.X%) |
| Partial Remission | XX (XX.X%) | XX (XX.X%) |
| Stable Disease | XX (XX.X%) | XX (XX.X%) |
| Progressive Disease | XX (XX.X%) | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) | XX (XX.X%) |
| ORR according to Lugano classification** | | |
| Patients with ORR | XX (XX.X%) | XX (XX.X%) |
| IC 95% for ORR rate | [XX.X% - XX.X%] | [XX.X% - XX.X%] |

Response of patients with no post-baseline response assessment (due to any reason) will be considered Not evaluated and patients will be considered non-responders.

Table 7.7-4 ORR\* evaluation - Confirmed cHL Set

| | Confirmed | cHL Set |
|---|---|---|
| | Cohort 1 | Cohort 2 |
| Best response according to Lugano classification* | | |
| Complete Response | XX (XX.X%) | XX (XX.X%) |
| Partial Remission | XX (XX.X%) | XX (XX.X%) |
| Stable Disease | XX (XX.X%) | XX (XX.X%) |
| Progressive Disease | XX (XX.X%) | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) | XX (XX.X%) |
| ORR according to Lugano classification** | | |
| Patients with ORR | XX (XX.X%) | XX (XX.X%) |
| IC 95% for ORR rate | [XX.X% - XX.X%] | [XX.X% - XX.X%] |

Response of patients with no post-baseline response assessment (due to any reason) will be considered Not evaluated and patients will be considered non-responders.

#### 7.7.2 Secondary efficacy endpoint analyses

### 7.7.2.1 Complete response rate

Table 7.7-5 CRR evaluation

| | Header |
|---------------------------------------------------|-----------------|
| Best response according to Lugano classification* | i |
| Complete Response | XX (XX.X%) |
| Partial Remission | XX (XX.X%) |
| Stable Disease | XX (XX.X%) |
| Progressive Disease | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| CRR according to Lugano classification** | |
| Patients with CRR | XX (XX.X%) |
| IC 95% for CRR rate | [XX.X% - XX.X%] |

Response of patients with no post-baseline response assessment (due to any reason) will be considered Not evaluated and patients will be considered non-responders.

<sup>\*</sup>Lugano classification: for each evaluation, metabolic response (PET-CT based) if available, radiologic response (CT-based) otherwise

<sup>\*\*</sup>ORR is defined as the proportion of patients who achieve a best response of CR or PR per the Lugano Classification (Cheson et al 2014) from the first dose of Tislelizumab until data cut or the start of a new anti-lymphoma therapy and determined by the investigator

<sup>\*</sup>Lugano classification: for each evaluation, metabolic response (PET-CT based) if available, radiologic response (CT-based) otherwise

<sup>\*\*</sup>ORR is defined as the proportion of patients who achieve a best response of CR or PR per the Lugano Classification (Cheson et al 2014) from the first dose of Tislelizumab until data cut or the start of a new anti-lymphoma therapy and determined by the investigator

<sup>\*</sup>Lugano classification: for each evaluation, metabolic response (PET-CT based) if available, radiologic response (CT-based) otherwise

<sup>\*\*</sup>CRR is defined as the proportion of patients who achieve a best response of CR per the Lugano Classification (Cheson et al 2014) from the first dose of Tislelizumab until data cut or the start of a new anti-lymphoma therapy and determined by the investigator

### 7.7.2.2 Duration of response

# 7.7.2.2.1 Duration of response events according to each censoring rule

Table 7.7-6 Events according to Duration of response definitions

| | Header |
|---|---|
| Patients with ORR as best response* | XXX |
| Event according to Duration of response definition with censoring on NALT | |
| No | XXX (XX.X%) |
| Yes | XXX (XX.X%) |
| If yes, type of event | |
| Progression/relapse | XXX (XX.X%) |
| Death from any cause | XXX (XX.X%) |
| Event according to Duration of response definition based on EMA censoring | |
| rules | |
| No | XXX (XX.X%) |
| Yes | XXX (XX.X%) |
| If yes, type of event | |
| Progression/relapse | XXX (XX.X%) |
| Death from any cause | XXX (XX.X%) |
| Event according to Duration of response definition with censoring on HSCT | |
| No . | XXX (XX.X%) |
| Yes | XXX (XX.X%) |
| If yes, type of event | ' ' |
| Progression/relapse | XXX (XX.X%) |
| Death from any cause | XXX (XX.X%) |

<sup>\*</sup>Lugano classification: for each evaluation, metabolic response (PET-CT based) if available, radiologic response (CT-based) otherwise, from the first dose of Tislelizumab until data cut or the start of a new anti-lymphoma therapy and determined by the investigator

#### 7.7.2.2.2 Main analysis: censoring on NALT

Table 7.7-7 Reasons for censoring DOR with censoring on NALT

| THE TOTAL PROPERTY OF THE DESCRIPTION OF THE DESCRI | on with tensoring on with |
|---|---|
| | Header |
| Censored patients | XXX (XX.X%) |
| Reason for Censoring | · |
| No event | XXX (XX.X%) |
| NALT without event | XXX (XX.X%) |
| NALT before progression or death | XXX (XX.X%) |

### Figure 7.7-1 Duration of response with censoring on NALT

Duration of response will be measured from the time of attainment of CR or PR to the date of first documented disease progression/relapse or death

Table 7.7-8 Duration of response with censoring on NALT -Survival Summary

| | Cohort | N | Number<br>of | Quartile | Estimate | 95% Cor<br>Inte | |
|---|---|---|---|---|---|---|---|
| | | | event | | | Lower | Upper |
| Duration of response (years) | Cohort 1 | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | Cohort 2 | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | Total Safety | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | Analysis Set | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |

Duration of response will be measured from the time of attainment of CR or PR to the date of first documented disease progression/relapse or death

Table 7.7-9 Duration of response with censoring on NALT — Survival Estimates

| THOSE 717 S DEFENDED OF TEST CONSTRUCTION OF THE DESCRIPTION | | | | | |
|---|---|---|---|---|---|
| Cohort | Time Point (years) | Duration of response | 95% Confide | ence Interval | Patients at risk |
| | | (%) | Lower | Upper | |
| Cohort 1 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Cohort 2 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Total Safety Analysis Set | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| | | 1 | | | |

Duration of response will be measured from the time of attainment of CR or PR to the date of first documented disease progression/relapse or death

### 7.7.2.2.3 Sensitivity analysis: censoring according to EMA censoring rules

### Figure 7.7-2 Duration of response according to EMA censoring rules

Duration of response will be measured from the time of attainment of CR or PR to the date of first documented disease progression/relapse or death

Table 7.7-10 Duration of response according to EMA censoring rules – Survival Summary

| table 7.7-10 Duration of response according to ENIA censoring rules—Survival Summary | | | | | | | |
|---|---|---|---|---|---|---|---|
| | Cohort | N | Number | Quartile | Estimate | 95% Cor | nfidence |
| | | | of | | | Inte | rval |
| | | | event | | | Lower | Upper |
| Duration of response | Cohort 1 | XX | XX | Q1 | XX.X | XX.X | XX.X |
| (years) | | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |

| Cohort 2 | XX | XX | Q1 | XX.X | XX.X | XX.X |
|---------------------------|----|----|--------|------|------|------|
| | | | Median | XX.X | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X | XX.X |
| Total Safety Analysis Set | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | | | Median | XX.X | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X | XX.X |

Duration of response will be measured from the time of attainment of CR or PR to the date of first documented disease progression/relapse or death

Table 7.7-11 Duration of response according to EMA censoring rules – Survival Estimates

| Table 7:7-11 Duration of response according to Liver censoring rules — But vival Estimates | | | | | |
|---|---|---|---|---|---|
| Cohort | Time Point (years) | Duration of response | 95% Confide | ence Interval | Patients at risk |
| | | (%) | Lower | Upper | |
| Cohort 1 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Cohort 2 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Total Safety Analysis Set | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |

Duration of response will be measured from the time of attainment of CR or PR to the date of first documented disease progression/relapse or death

#### 7.7.2.2.4 Sensitivity analysis: censoring on HSCT only

Table 7.7-12 Reasons for censoring DOR with censoring on HSCT

| the fif 12 Reasons for consoring D of the consoring of 115 c | |
|---|---|
| | Header |
| Censored patients | XXX (XX.X%) |
| Reason for Censoring | |
| No event | XXX (XX.X%) |
| HSCT without event | XXX (XX.X%) |
| HSCT before progression or death | XXX (XX.X%) |

### Figure 7.7-3 Duration of response with censoring on HSCT

Duration of response will be measured from the time of attainment of CR or PR to the date of first documented disease progression/relapse or death

Table 7.7-13 Duration of response with censoring on HSCT –Survival Summary

| Table 7.7-13 Dulation of i | <u>гезропзе wit</u> | <u>п сепз</u> | <u>отния оп</u> | <u> 1 11 501 - 501 </u> | <u>vivai Summai y</u> | | |
|---|---|---|---|---|---|---|---|
| | Cohort | N | Number | Quartile | Estimate | 95% Cor | nfidence |
| | | | of | | | Inte | rval |
| | | | event | | | Lower | Upper |
| Duration of response (years) | Cohort 1 | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | Cohort 2 | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | Total | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | Safety | | | Median | XX.X | XX.X | XX.X |
| | Analysis | | | Q3 | XX.X | XX.X | XX.X |
| | Set | | | | | | 1 |

Duration of response will be measured from the time of attainment of CR or PR to the date of first documented disease progression/relapse or death

<u>Table 7.7-14 Duration of response with censoring on HSCT-Survival Estimates</u>

| Cohort Time Point (years) 95% Confidence Interval Patients at risk |
|--------------------------------------------------------------------------|
|--------------------------------------------------------------------------|

### TIRHOL - Statistical Analysis Plan


| | | Duration of response | Lower | Upper | |
|---------------------------|---|----------------------|-------|-------|----|
| | | (%) | | | |
| Cohort 1 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Cohort 2 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Total Safety Analysis Set | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |

Duration of response will be measured from the time of attainment of CR or PR to the date of first documented disease progression/relapse or death

### 7.7.2.3 Time to response

Table 7.7-15 Time to response

| Table 7.7 15 Time to response | |
|-------------------------------|--------------|
| | Header |
| Patients with ORR as best | XXX |
| response* | |
| Time to response (months) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |

<sup>\*</sup>Lugano classification: for each evaluation, metabolic response (PET-CT based) if available, radiologic response (CT-based) otherwise, from the first dose of Tislelizumab until data cut or the start of a new anti-lymphoma therapy and determined by the investigator

### 7.7.3 Exploratory endpoint analyses

7.7.3.1 Progression free survival (PFS)

### 7.7.3.1.1 PFS events according to each censoring rule

Table 7.7-16 Events according to PFS definitions

| | Header |
|---|---|
| Event according PFS definition with censoring on NALT | |
| No | XXX (XX.X%) |
| Yes | XXX (XX.X%) |
| If yes, type of event | 7000 (700,775) |
| Progression/relapse | XXX (XX.X%) |
| Death from any cause | XXX (XX.X%) |
| Event according to PFS definition based on EMA censoring rules | |
| No | XXX (XX.X%) |
| Yes | XXX (XX.X%) |
| If yes, type of event | |
| Progression/relapse | XXX (XX.X%) |
| Death from any cause | XXX (XX.X%) |
| Event according to PFS definition with censoring on HSCT | |
| No | XXX (XX.X%) |
| Yes | XXX (XX.X%) |
| If yes, type of event | |
| Progression/relapse | XXX (XX.X%) |
| Death from any cause | XXX (XX.X%) |

<sup>\*</sup>Lugano classification: for each evaluation, metabolic response (PET-CT based) if available, radiologic response (CT-based) otherwise, from the first dose of Tislelizumab until data cut or the start of a new anti-lymphoma therapy and determined by the investigator

### 7.7.3.1.2 Main analysis: censoring on NALT

Table 7.7-17 Reasons for censoring PFS with censoring on NALT

| _ | Header |
|---------------------------------------|-------------|
| Censored patients | XXX (XX.X%) |
| Reason for Censoring | · |
| No event | XXX (XX.X%) |
| NALT without event | XXX (XX.X%) |
| NALT before progression or death | XXX (XX.X%) |
| No baseline reviewed tumor assessment | XXX (XX.X%) |

### Figure 7.7-4 PFS with censoring on NALT

<u>Table 7.7-18 PFS with censoring on NALT – Survival Summary</u>

| | Cohort | N | Number | Quartile | Estimate | | nfidence |
|---|---|---|---|---|---|---|---|
| | | | of | | | Inte | erval |
| | | | event | | | Lower | Upper |
| PFS (years) | Cohort 1 | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | Cohort 2 | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | | XX | XX | Q1 | XX.X | XX.X | XX.X |

| Total Safety | Median | XX.X | XX.X | XX.X |
|--------------|--------|------|------|------|
| Analysis Set | Q3 | XX.X | XX.X | XX.X |

Table 7.7-19 PFS with censoring on NALT - Survival Estimates

| THOIC / // IN II S II IN | COMPOSITION OF THE | LLI SULTINILES | *************************************** | | |
|---|---|---|---|---|---|
| Cohort | Time Point (years) | PFS (%) | 95% Confid | dence Limits | Patients at risk |
| | | | Lower | Upper | |
| Cohort 1 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Cohort 2 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Total Safety Analysis Set | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |

# 7.7.3.1.3 Sensitivity analysis: censoring according to EMA censoring rules

### Figure 7.7-5 PFS with censoring according to EMA censoring rules

Table 7.7-20 PFS with censoring according to EMA censoring rules – Survival Summary

| Table 7.7-20 IIS With te | nooring according | to Livi | 21 CCH50 | III I tales = | ui (I) ui Summi | <u> , </u> | |
|---|---|---|---|---|---|---|---|
| | Cohort | N | Number | Quartile | Estimate | 95% Co | nfidence |
| | | | of | | | Inte | rval |
| | | | event | | | Lower | Upper |
| PFS (years) | Cohort 1 | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | Cohort 2 | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | Total Safety | | | Median | XX.X | XX.X | XX.X |
| | Analysis Set | | | Q3 | XX.X | XX.X | XX.X |

Table 7.7-21 PFS with censoring according to EMA censoring rules—Survival Estimates

| Table 7.7-21 TTS With | CCHSOTINE MCCOL | WILL TO LIVING COMP | JIIII I WILL | , Starting | di Liberinitetos |
|---|---|---|---|---|---|
| Cohort | Time Point (years) | PFS (%) | 95% Confid | lence Limits | Patients at risk |
| | | | Lower | Upper | |
| Cohort 1 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Cohort 2 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| Total Safety Analysis Set | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |

### 7.7.3.1.4 Sensitivity analysis: censoring on HSCT

### Table 7.7-22 Reasons for censoring PFS with censoring on HSCT

### TIRHOL - Statistical Analysis Plan


| | Header |
|---------------------------------------|-------------|
| Censored patients | XXX (XX.X%) |
| Reason for Censoring | |
| No event | XXX (XX.X%) |
| HSCT without event | XXX (XX.X%) |
| HSCT before progression or death | XXX (XX.X%) |
| No baseline reviewed tumor assessment | XXX (XX.X%) |

# Figure 7.7-6 PFS with censoring on HSCT

Table 7.7-23 PFS with censoring on HSCT - Survival Summary

| | Cohort | N | Number | Quartile | Estimate | 95% Cor | nfidence |
|---|---|---|---|---|---|---|---|
| | | | of | | | Inte | rval |
| | | | event | | | Lower | Upper |
| PFS (years) | Cohort 1 | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | Cohort 2 | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | Total Safety | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | Analysis Set | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |

Table 7.7-24 PFS with censoring on HSCT - Survival Estimates

| Table 7.7-24 1 F5 with censoring on 115c1 - Survival Estimates | | | | | |
|---|---|---|---|---|---|
| Cohort | Time Point (years) | me Point (years) PFS (%) 95% Confidence Limit | | lence Limits | Patients at risk |
| | | | Lower | Upper | |
| Cohort 1 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Cohort 2 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| | 0 | XX.X | XX.X | XX.X | XX |
| Total Safety Analysis Set | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |

# 7.7.3.2 Overall survival (OS)

Table 7.7-25 Events according to OS definition

| Table 7.7-23 Events according to OS definition | |
|---|---|
| | Header |
| Event according OS definition | |
| No | XXX (XX.X%) |
| Yes | XXX (XX.X%) |

# **Figure 7.7-7 OS**

Table 7.7-26 OS – Survival Summary

| | Cohort | N | Number | Quartile | Estimate | 95% Coi | nfidence |
|---|---|---|---|---|---|---|---|
| | | | of | | | Interval | |
| | | | event | | | Lower | Upper |
| OS (years) | Cohort 1 | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | Cohort 2 | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |
| | Total Safety | XX | XX | Q1 | XX.X | XX.X | XX.X |
| | Analysis Set | | | Median | XX.X | XX.X | XX.X |
| | | | | Q3 | XX.X | XX.X | XX.X |

Table 7.7-27 OS – Survival Estimates

| Tubic 7.7 27 Ob Bul | vivai Listimates | | | | |
|---|---|---|---|---|---|
| Cohort | Time Point (years) | OS (%) | 95% Confidence Limits | | Patients at risk |
| | | | Lower | Upper | |
| Cohort 1 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Cohort 2 | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |
| Total Safety Analysis Set | 0 | XX.X | XX.X | XX.X | XX |
| | 1 | XX.X | XX.X | XX.X | XX |
| | 2 | XX.X | XX.X | XX.X | XX |
| | | XX.X | XX.X | XX.X | XX |

# 7.7.4 Progression / Relapse

7.7.4.1 Patients presenting with progression/relapse

Table 7.7-28 Patients presenting with progression/relapse

| | Header |
|---------------------------------|------------|
| Progression/Relapse | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, initial involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, new involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, nodal involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, extra-nodal involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

### 7.7.4.2 Progression/relapse documentation

Table 7.7-29 Progression/relapse documentation

| | Header |
|----------------------------|------------|
| Histological documentation | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Cytological documentation | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

Note: N corresponds to patients presenting with progression

### 7.7.4.3 New anti-cancer therapy for progression/relapse

Table 7.7-30 New anti-cancer therapy for progression/relapse

| Table 7.7-30 New anti-cancer therapy for pro | |
|----------------------------------------------|------------|
| | Header |
| Progression/relapse treatment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Monoclonal antibody | , , , |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Other immunotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Chemotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Radiotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Autologous transplant | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Allogenic transplant | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| IMiD agents | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Epigenetic modifiers agents | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Kinase inhibitor | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Other anti-cancer therapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

Note: N corresponds to patients presenting with progression

# <u>Listing 7.7-3 Patients with monoclonal antibody therapy as progression/relapse treatment - Safety</u>

Analysis Set (XX patients) Cohort Patient Date of Drug(s) name of Start date of End date of Date of Monoclonal identification monoclonal progression / monoclonal monoclonal antibody first dose number antibody antibody antibody relapse Yes Χ X Χ

# Listing 7.7-4 Patients with other immunotherapy as progression/relapse treatment - Safety Analysis Set

| (XX patients | <u>)</u> | | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of first dose | Date of<br>progression /<br>relapse | Other immunotherapy | Drug(s) name of<br>other<br>immunotherapy | Start date of<br>other<br>immunotherapy | End date of other immunotherapy |
| X | | | | Yes | | | |


# <u>Listing 7.7-5 Patients with chemotherapy as progression/relapse treatment – Safety Analysis Set (XX</u>

| <u>patients)</u> | | | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of first dose | Date of<br>progression /<br>relapse | Chemotherapy | Drug(s) name of<br>chemotherapy | Start date of<br>chemotherapy | End date of<br>chemotherapy |
| X | | | | Yes | | | |

### Listing 7.7-6 Patients with radiotherapy as progression/relapse treatment - Safety Analysis Set (XX

| <u>patients)</u> | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of first dose | Date of<br>progression /<br>relapse | Radiotherapy | Anatomic site of radiotherapy | Dose of<br>radiotherapy<br>(Gy) | Start date of radiotherapy | End date of radiotherapy |
| X | | | | Yes | | | | |

### <u>Listing 7.7-7 Patients with autologous transplant as progression/relapse treatment – Safety Analysis Set</u>

| (XX patients | <u></u> | | | | | |
|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of<br>first dose | Date of<br>progression /<br>relapse | Autologous<br>transplant | Autologous<br>transplant<br>conditioning<br>regimen before<br>HSCT | Date of<br>autologous<br>transplant |
| X | | | | Yes | | |

### <u>Listing 7.7-8 Patients with allogenic transplant as progression/relapse treatment - Safety Analysis Set</u>

| (XX patients) | ) | | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of first dose | Date of<br>progression /<br>relapse | Allogenic<br>transplant | Allogenic<br>transplant<br>conditioning<br>regimen before<br>HSCT | Type of<br>allogenic<br>transplant | Date of<br>allogenic<br>transplant |
| X | | | | Yes | | | |

# <u>Listing 7.7-9 Patients with IMiD agents as progression/relapse treatment - Safety Analysis Set (XX</u>

| <u>patients)</u> | | | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of<br>first dose | Date of<br>progression /<br>relapse | Allogenic<br>transplant | Allogenic<br>transplant<br>conditioning<br>regimen before<br>HSCT | Type of<br>allogenic<br>transplant | Date of<br>allogenic<br>transplant |
| X | | | | Yes | | | |

### <u>Listing 7.7-10 Patients with epigenetic modifiers agents as progression/relapse treatment - Safety</u>

| Analysis Set | (XX patients) | ) | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of first dose | Date of progression / relapse | Epigenetic<br>modifiers agents | Drug(s) name of<br>epigenetic<br>modifiers agents | Start date of<br>epigenetic<br>modifiers agents | End date of<br>epigenetic<br>modifiers<br>agents |
| X | | | | Yes | | | |

# <u>Listing 7.7-11 Patients with kinase inhibitor as progression/relapse treatment – Safety Analysis Set (XX</u>

| <u>patients)</u> | | | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of first dose | Date of progression / relapse | Epigenetic<br>modifiers agents | Drug(s) name of<br>epigenetic<br>modifiers agents | Start date of<br>epigenetic<br>modifiers agents | End date of<br>epigenetic<br>modifiers<br>agents |
| X | | | | Yes | | | |

# <u>Listing 7.7-12 Patients with Other anti-cancer therapy as progression/relapse treatment - Safety Analysis Set (XX patients)</u>

### TIRHOL - Statistical Analysis Plan


| Cohort | Patient<br>identification<br>number | Date of<br>first dose | Date of progression / relapse | Other anti-<br>cancer therapy | Drug(s) name of<br>other anti-<br>cancer therapy | Start date of<br>other anti-<br>cancer therapy | End date of<br>other anti-<br>cancer<br>therapy |
|---|---|---|---|---|---|---|---|
| X | | | | Yes | | | |

### 7.7.4.4 Response after additional treatment(s)

Table 7.7-31 Response after additional treatment(s)

| Table 7.7-51 Response after addition | nai ti catincitys) |
|--------------------------------------|--------------------|
| | Header |
| If progression/relapse, Response at | ter additional |
| treatment(s) | |
| Complete Response | XX (XX.X%) |
| Partial Response | XX (XX.X%) |
| Stable Disease | XX (XX.X%) |
| Progressive Disease | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Missing | xx (xx.x%) |

Note: N corresponds to patients presenting with progression/relapse

# 7.7.5 New anti-cancer therapy given prior to disease progression

Table 7.7-32 New anti-cancer therapy given prior to progression/relapse

| | Header |
|----------------------------------------|------------|
| New anti-cancer therapy given prior to | |
| progression/relapse | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Monoclonal antibody | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Other immunotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Chemotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Radiotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Autologous transplant | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Allogenic transplant | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| IMiD agents | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Epigenetic modifiers agents | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Kinase inhibitor | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Other anti-cancer therapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

Note: N corresponds to patients presenting with progression

# Listing 7.7-13 Patients with monoclonal antibody therapy given prior to progression/relapse treatment

| - Safety | Analy | vsis S | et (XX | X patients) | ) |
|----------|-------|--------|--------|-------------|---|

| Cohe | ort | Patient<br>identification<br>number | Date of first dose | Date of<br>progression /<br>relapse | Monoclonal<br>antibody | Drug(s) name of<br>monoclonal<br>antibody | Start date of<br>monoclonal<br>antibody | End date of<br>monoclonal<br>antibody |
|---|---|---|---|---|---|---|---|---|
| X | | | | | Yes | | | |

### <u>Listing 7.7-14 Patients with other immunotherapy given prior to progression/relapse treatment - Safety</u>

| Analysis Set | (XX patients | <u>s)</u> | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of first dose | Date of<br>progression /<br>relapse | Other<br>immunotherapy | Drug(s) name of<br>other<br>immunotherapy | Start date of<br>other<br>immunotherapy | End date of other immunotherapy |
| X | | | | Yes | | | |

# <u>Listing 7.7-15 Patients with chemotherapy given prior to progression/relapse treatment - Safety</u>

| <u>Analysis Set (</u> | (XX patients) | | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of first dose | Date of<br>progression /<br>relapse | Chemotherapy | Drug(s) name of<br>chemotherapy | Start date of<br>chemotherapy | End date of<br>chemotherapy |
| X | | | | Yes | | | |

# Listing 7.7-16 Patients with radiotherapy given prior to progression/relapse treatment – Safety Analysis

| Set (XX pation | ents) | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of first dose | Date of<br>progression /<br>relapse | Radiotherapy | Anatomic site of radiotherapy | Dose of<br>radiotherapy<br>(Gy) | Start date of radiotherapy | End date of radiotherapy |
| X | | | | Yes | | | | |

### Listing 7.7-17 Patients with autologous transplant given prior to progression/relapse treatment – Safety

| <u>Analysis Set</u> | (XX patients | | |
|---------------------|---------------------------|---------|------|
| Cohort | | | |
| | Patient<br>identification | Date of | Drog |

| Cohort | Patient<br>identification<br>number | Date of first dose | Date of<br>progression /<br>relapse | Autologous<br>transplant | Autologous<br>transplant<br>conditioning<br>regimen before<br>HSCT | Date of<br>autologous<br>transplant |
|---|---|---|---|---|---|---|
| X | | | | Yes | | |

# <u>Listing 7.7-18 Patients with allogenic transplant given prior to progression/relapse treatment - Safety</u>

Analysis Set (XX natients)

| Anarysis Sct | (2X2X patients | L | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of<br>first dose | Date of<br>progression /<br>relapse | Allogenic<br>transplant | Allogenic<br>transplant<br>conditioning<br>regimen before<br>HSCT | Type of<br>allogenic<br>transplant | Date of<br>allogenic<br>transplant |
| X | | | | Yes | | | |

# Listing 7.7-19 Patients with IMiD agents given prior to progression/relapse treatment – Safety Analysis

| SCI (AA PAH | <u>спіз)</u> | | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of<br>first dose | Date of<br>progression /<br>relapse | Allogenic<br>transplant | Allogenic<br>transplant<br>conditioning<br>regimen before<br>HSCT | Type of<br>allogenic<br>transplant | Date of<br>allogenic<br>transplant |
| X | | | | Yes | | | |

# Listing 7.7-20 Patients with epigenetic modifiers agents given prior to progression/relapse treatment -

Safety Analysis Set (XX patients) Cohort End date of Patient Date of Drug(s) name of Start date of Date of **Epigenetic** epigenetic identification epigenetic epigenetic progression / modifiers first dose modifiers agents number relapse modifiers agents modifiers agents agents Χ Yes

# Listing 7.7-21 Patients with kinase inhibitor given prior to progression/relapse treatment — Safety

| <u>Analysis Set</u> | (XX patients) | <u>)</u> | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of first dose | Date of progression / relapse | Epigenetic<br>modifiers agents | Drug(s) name of<br>epigenetic<br>modifiers agents | Start date of<br>epigenetic<br>modifiers agents | End date of<br>epigenetic<br>modifiers<br>agents |
| X | | | | Yes | | | |

### <u>Listing 7.7-22 Patients with Other anti-cancer therapy given prior to progression/relapse treatment —</u>

| Safety Analy | sis Set (XX p | <u>atients)</u> | | | | | |
|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>identification<br>number | Date of first dose | Date of progression / relapse | Other anti-<br>cancer therapy | Drug(s) name of<br>other anti-<br>cancer therapy | Start date of<br>other anti-<br>cancer therapy | End date of<br>other anti-<br>cancer<br>therapy |
| X | | | | Yes | | | |

# 7.8 Extent of exposure

### **7.8.1** Cycles

Table 7.8-1 Treatment durations

| | Header |
|--------------------------------------------|--------------|
| Duration of Tislelizumab treatment (weeks) | |
| N | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |

The duration of Tislelizumab treatment (weeks) is calculated as (date of last dose + 21 days - date of first dose)/7

Table 7.8-2 Tislelizumab cycles administered

| | Header |
|---------------------------|--------------|
| Cycles performed | |
| Cycle 1 | XX (XX.X%) |
| Cycle 2 | XX (XX.X%) |
| ••• | XX (XX.X%) |
| Number of cycles received | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |

EN-SOP-ST-03-Temp-01-SAP Template (Phase II/III) - V2.0 - Effective date: 14/12/2016

### 7.8.2 Dose

Table 7.8-3 Tislelizumab exposure

| 1 abie 7.6-3 Tisienzumab exposure | Header |
|-------------------------------------------------|--------------|
| | ricadei |
| Cumulative total dose received per patient (mg) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |
| Dose intensity (mg/day)* | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |
| Relative dose intensity** | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| <75% | XX (XX.X%) |
| [75%-90%[ | XX (XX.X%) |
| [90%-110%[ | XX (XX.X%) |
| [110%-125%[ | XX (XX.X%) |
| >=125% | XX (XX.X%) |

<sup>\*</sup> Dose intensity is defined as:

Cumulative total dose received / duration of treatment in days

Dose intensity/Planned dose intensity

Planned dose intensity = 200mg/21 days

<sup>\*\*</sup> Relative dose intensity is defined as:

### 7.8.3 Dose modifications

Table 7.8-4 Modifications of scheduled Tislelizumab infusion by patient

| | Header |
|----------------------------------------|------------|
| At least one modification of scheduled | ĺ |
| Tislelizumab infusion | |
| Yes | XX (XX.X%) |
| No | XX (XX.X%) |
| If yes, type of modification* | |
| Drug withdrawn | XX (XX.X%) |
| Drug interrupted at least once | XX (XX.X%) |
| Drug delayed at least once | XX (XX.X%) |
| Cycle of drug withdraw | |
| 1 | XX (XX.X%) |
| | XX (XX.X%) |
| Patients with drug interruption | XX |
| Number of drug interruptions | |
| 1 | XX (XX.X%) |
| | XX (XX.X%) |
| First cycle with drug interruption | |
| 1 | XX (XX.X%) |
| | XX (XX.X%) |
| Patients with drug delay | XX |
| Number of drug delays | |
| 1 | XX (XX.X%) |
| | XX (XX.X%) |
| First cycle with drug delay | |
| 1 | XX (XX.X%) |
| | XX (XX.X%) |

N=Number of patients

Table 7.8-5 Modifications of scheduled Tislelizumab infusion by modification

| | Header |
|-----------------------------|------------|
| Type of modification | |
| Drug withdrawn | XX (XX.X%) |
| Drug interrupted | XX (XX.X%) |
| Drug delayed | XX (XX.X%) |
| If drug withdrawn, reason | |
| AE | XX (XX.X%) |
| Other | XX (XX.X%) |
| If other, specify | |
| | XX (XX.X%) |
| If drug interrupted, reason | |
| AE | XX (XX.X%) |
| Other | XX (XX.X%) |
| If other, specify | |
| | XX (XX.X%) |
| If drug delayed, reason | ' ' |
| AE | XX (XX.X%) |
| Other | XX (XX.X%) |
| If other, specify | ' ' |
| | XX (XX.X%) |

N=Number of dose modifications (up to 3 dose modifications may be reported by cycle)

<sup>\*</sup> The sum of types of modification can be > 100% because the types are not mutually exclusive

Table 7.8-6 Modifications of scheduled Tislelizumab infusion by cycle in cohort 1

| | Coho | rt X |
|------------------------------|------------|------------|
| | Cycle 1 | Cyde |
| | N=XX | N=XX |
| Type of modification* | | |
| Drug withdrawn | XX (XX.X%) | XX (XX.X%) |
| Drug interrupted | XX (XX.X%) | XX (XX.X%) |
| Drug delayed | XX (XX.X%) | XX (XX.X%) |
| If drug withdrawn, reason | | |
| AE | XX (XX.X%) | XX (XX.X%) |
| Other | XX (XX.X%) | XX (XX.X%) |
| If drug interrupted, reason | | |
| AE | XX (XX.X%) | XX (XX.X%) |
| Other | XX (XX.X%) | XX (XX.X%) |
| If drug delayed, reason** | | |
| AE | XX (XX.X%) | XX (XX.X%) |
| Other | XX (XX.X%) | XX (XX.X%) |
| Number of dose interruptions | | · · · |
| 0 | XX (XX.X%) | XX (XX.X%) |
| 1 | XX (XX.X%) | XX (XX.X%) |
| 2 | XX (XX.X%) | XX (XX.X%) |
| 3 | XX (XX.X%) | XX (XX.X%) |
| Number of dose delays | | |
| 0 | XX (XX.X%) | XX (XX.X%) |
| 1 | XX (XX.X%) | XX (XX.X%) |
| 2 | XX (XX.X%) | XX (XX.X%) |
| 3 | XX (XX.X%) | XX (XX.X%) |

N=Number of patients with the cycle performed

Table 7.8-7 Modifications of scheduled Tislelizumab infusion by cycle in cohort 2

<sup>\*</sup> The sum can be >100% because the types are not mutually exclusive

<sup>\*\*</sup> The sum can be >100% because up to 3 modifications by cycle

Listing 7.8-1 Drug withdrawn due to AE - Safety Analysis Set (XX drug withdrawn reported by XX patients)

| L15ting /.o-1 1 | Ji ug withulan | II UU | t to AL - | - Saicty A | Halysis SC | t (AA urug | withuraw. | птср | or ica by 2 | <b>3.</b> 7. 10 pa | <u>исиіз)</u> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort | Patient | Sex | Age | Date of | Number of | Drug wi | Adverse Event | | | | | | | | | |
| | Identification | | (years) | first dose | cycles | | | | Onset | End | Date when AE | Intensity | Highest | Tisleliz | umab | Outcome |
| | Number | | | | received | | | | date | date became at onset intensity | | | | | | |
| | | | | | | | | | | | serious | date | | | | |
| | | | | | | Cycle of | Reason of | | | | | | | Relation- | Action | |
| | | | | | | drug | drug | | | | | | | ship | taken | |
| | | | | | | withdrawal | withdrawal | | | | | | | | | |
| X | XX | X | XX | XX/XX/XX | X | X | XX | XX | XX/XX/XX | XX/X | XX/XX/XXXX | X | X | X | XX | X |
| | | | | XX | | | | | XX | X/XX | | | | | | |
| | | | | | | | | | | XX | | | | | | |

Listing 7.8-2 Drug interrupted due to AE - Safety Analysis Set (XX drug interrupted reported by XX patients)

| - | LISHING 7.0-2 D | <u>n ug mierrupi</u> | <del>cu uu</del> | t to AL | - Saicty A | mary sis so | ti (AA uru | g micrrupi | cuic | JOI ICU DY | $\Lambda\Lambda$ | <u>atients)</u> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Cohort | Patient | Sex | Age | Date of | Number of | Dr | Adverse Event | | | | | | | | | |
| | | Identification | | (years) | first dose | cycles | interruption | | PT | PT Onset End Date when AE Intensity Highest Tislelizuma | | umab | Outcome | | | | |
| | | Number | | | | received | | | | date | date | ate became at onset intensity | | | | | |
| | | | | | | | | | | | | serious | date | | | | |
| | | | | | | | Cycle of | Reason of | | | | | | | Relation- | Action | |
| | | | | | | | drug | drug | | | | | | | ship | taken | |
| | | | | | | | interruption | interruption | | | | | | | | | |
| | X | XX | X | XX | XX/XX/XX | X | X | XX | XX | XX/XX/XX | XX/X | XX/XX/XXXX | X | X | X | XX | X |
| | | | | | XX | | | | | XX | X/XX | | | | | | |
| | | | | | | | | | | | XX | | | | | | |

Listing 7.8-3 Drug delayed due to AE - Safety Analysis Set (XX drug delayed reported by XX patients)

| Cohort | Patient | Sex | Age | Date of | Number of | Drug | | Adverse Event | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Identification | | (years) | first dose | cycles | delay | | delay | | PT | Onset | End | Date when AE | Intensity | Highest | Tisleliz | umab | Outcome |
| | Number | | | | received | | • | | date | date | ate became at onset intensity | | | | | | | |
| | | | | | | | | | | | serious | date | | | | | | |
| | | | | | | Cycle of | Reason of | | | | | | | Relation- | Action | | | |
| | | | | | | drug delay | drug delay | | | | | | | ship | taken | | | |
| X | XX | X | XX | XX/XX/XX | X | X | XX | XX | XX/XX/XX | XX/X | XX/XX/XXXX | X | X | X | XX | X | | |
| | | | | XX | | | | | XX | X/XX | | | | | | | | |
| | | | | | | | | | | XX | | | | | | | | |

# 7.9 Safety analysis

# 7.9.1 Treatment Emergent Adverse Events

7.9.1.1 Summary

**Table 7.9-1 Overview of Treatment Emergent Adverse Events** 

| Table 7.5 1 Overview of Treatment Emergent Maverse Events | |
|---|---|
| | Header |
| Patients with at least one TEAE | XX (XX.X%) |
| If so, number of TEAEs by patient | |
| Number | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |
| Patients with at least one TEAE with grade >= 3 | XX (XX.X%) |
| Patients with at least one serious TEAE | XX (XX.X%) |
| Patients with at least one TEAE leading to discontinuation or interruption of Tislelizumab | XX (XX.X%) |
| Patients with at least one serious TEAE leading to discontinuation or interruption of Tislelizumab | XX (XX.X%) |
| Patients with at least one fatal TEAE | XX (XX.X%) |
| Patients with at least one irAE (BG charter) | XX (XX.X%) |
| Patients with at least one other malignancy* | XX (XX.X%) |

<sup>\*</sup> Per other primary malignancy page

**Table 7.9-2 Characteristics of Treatment Emergent Adverse Events** 

| | Header |
|--------------------------------------|---------------|
| TFAF Serious | |
| No. | XX (XX.X%) |
| Yes | XX (XX.X%) |
| TEAE onset Intensity | // (//.// //) |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| 4 | XX (XX.X%) |
| 5 | XX (XX.X%) |
| TEAE highest Intensity | |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 2 3 | XX (XX.X%) |
| 4 | XX (XX.X%) |
| 5 | XX (XX.X%) |
| Relationship with Tislelizumab | |
| Related | XX (XX.X%) |
| Unrelated | XX (XX.X%) |
| Action taken with Tislelizumab | |
| Permanent stop | XX (XX.X%) |
| Temporarily stop | XX (XX.X%) |
| Dose adaptation | XX (XX.X%) |
| Unchanged | XX (XX.X%) |
| Temporarily stop and Dose adaptation | XX (XX.X%) |
| Outcome | |
| Not recovered/Not resolved | XX (XX.X%) |
| Recovered/Resolved | XX (XX.X%) |
| Recovered/Resolved with sequelae | XX (XX.X%) |
| Death | XX (XX.X%) |
| Unknown | XX (XX.X%) |
| AESI | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

# 7.9.1.2 Treatment emergent adverse events (TEAEs)

# Table 7.9-3 Description of TEAEs by SOC/PT

| System<br>Preferred Term | Organ | Class | Header | | |
|---|---|---|---|---|---|
| | | | F | Patients | Events |
| TEAE | | | XX | (XX.X%) | XX |
| SOC1 | | | XX | (XX.X%) | XX |
| PT1 | | | XX | (XX.X%) | XX |
| PT2 | | | XX | (XX.X%) | XX |
| | | | XX | (XX.X%) | XX |
| SOC2 | | | XX | (XX.X%) | XX |
| PT1 | | | XX | (XX.X%) | XX |
| PT2 | | | XX | (XX.X%) | XX |
| | | | XX | (XX.X%) | l xx |

Table 7.9-4 Description of TEAEs by highest grade and SOC/PT - Cohort 1

| System Organ<br>Class | | | | | | | Safety A | nalysis Set - (<br>N=XX | Cohort 2 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | | Grade 1 | | | Grade 2 | | | Grade 3 | | | Grade 4 | | | | |
| | | | | Patients Events Patients Events Events Events | | | | Patients | | Events | Pá | atients | Events | | |
| TEAE | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| SOC1 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| SOC2 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |

# Table 7.9-5 Description of TEAEs by highest grade and SOC/PT - Cohort 2

### 7.9.1.3 Grade 3 and above TEAEs

Table 7.9-6 Description of TEAEs with highest grade >=3 by SOC/PT

| System | Organ | Class | | Header | |
|-----------------|-------|-------|-------------|---------|----|
| Preferred Term | | | Patients Ev | | |
| TEAE with grade | >=3 | | XX | (XX.X%) | XX |
| SOC1 | | | XX | (XX.X%) | XX |
| PT1 | | | XX | (XX.X%) | XX |
| PT2 | | | XX | (XX.X%) | XX |
| | | | XX | (XX.X%) | XX |
| SOC2 | | | XX | (XX.X%) | XX |
| PT1 | | | XX | (XX.X%) | XX |
| PT2 | | | XX | (XX.X%) | XX |
| | | | XX | (XX.X%) | XX |

### 7.9.1.4 Treatment-related TEAEs

# Table 7.9-7 Description of treatment-related TEAEs by SOC/PT

| System 0 Preferred Term | organ Class | | Header | |
|-------------------------|---------------------|----|----------|----|
| Treferred Term | | F | Patients | |
| Treatment-related TEAE | ntment-related TEAE | | | |
| SOC1 | | XX | (XX.X%) | XX |
| PT1 | | XX | (XX.X%) | XX |
| PT2 | | XX | (XX.X%) | XX |
| | | XX | (XX.X%) | XX |
| SOC2 | | XX | (XX.X%) | XX |
| PT1 | | XX | (XX.X%) | XX |
| PT2 | | XX | (XX.X%) | XX |
| | | XX | (XX.X%) | XX |

Table 7.9-8 Description of treatment-related TEAEs by highest grade and SOC/PT - Cohort 1

| Tuble 7.5 0 Desci | able 7.5-0 Description of treatment-related TEAEs by mightest grade and 50c/11 - Conort 1 | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ | | | | | | | Safety A | nalysis Set - ( | Cohort 1 | | | | | | |
| Class | | | | | | | | N=XX | | | | | | | |
| Preferred Term | Grade 1 | | | Grade 2 Grade 3 | | | | | | Grade 4 | | Grade 5 | | | |
| | Patients Events | | | Pa | atients | Events | s Patients Events | | | P | atients | Events | Pa | atients | Events |
| Treatment-related | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| TEAE | | | | | | | | | | | | | | | |
| SOC1 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| SOC2 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |

Table 7.9-9 Description of treatment-related TEAEs by highest grade and SOC/PT - Cohort 2

7.9.1.5 Treatment-related TEAEs with Grade 3 or above

Table 7.9-10 Description of treatment-related TEAEs with highest grade >= 3 by SOC/PT

| System | Organ | Class | | Header | |
|------------------|-----------------------|-------|----|----------|--------|
| Preferred Term | | | F | Patients | Events |
| Treatment-relate | d TEAE with grade >=3 | | XX | (XX.X%) | XX |
| SOC1 | | | XX | (XX.X%) | XX |
| PT1 | | | XX | (XX.X%) | XX |
| PT2 | | | XX | (XX.X%) | XX |
| | | | XX | (XX.X%) | XX |
| SOC2 | | | XX | (XX.X%) | XX |
| PT1 | | | XX | (XX.X%) | XX |
| PT2 | | | XX | (XX.X%) | XX |
| | | | XX | (XX.X%) | XX |

7.9.1.6 TEAEs leading to discontinuation or interruption of study treatment

Table 7.9-11 Description of TEAEs leading to discontinuation or interruption of Tislelizumab by SOC/PT

| System | Organ | Class | | | |
|---|---|---|---|---|---|
| Preferred Term | | P | atients | Events | |
| TEAE leading to dis<br>Tislelizumab | scontinuation or interruption of | | XX | (XX.X%) | ХХ |
| SOC1 | | | XX | (XX.X%) | XX |
| PT1 | | | XX | (XX.X%) | XX |
| PT2 | | | XX | (XX.X%) | XX |
| | | | XX | (XX.X%) | XX |
| SOC2 | | | XX | (XX.X%) | XX |

# TIRHOL - Statistical Analysis Plan

### Version 1.0 – 12APR2023

| System | Organ | Class | | | |
|----------------|-------|-------|----|--------------|----|
| Preferred Term | | | P | Patients Eve | |
| PT1 | | | XX | (XX.X%) | XX |
| PT2 | | | XX | (XX.X%) | XX |
| | | | XX | (XX.X%) | XX |

### 7.9.1.7 Fatal events

Table 7.9-12 Description of fatalFatal\* AEs by SOC/PT

| System Organ Class<br>Preferred Term | | Header | |
|--------------------------------------|-----|----------|----|
| | T I | Patients | |
| Fatal AE | XX | (XX.X%) | XX |
| SOC1 | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX |
| SOC2 | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX |

<sup>\*</sup>Fatal AE are TEAE of grade 5

Listing 7.9-1 Fatal\* AEs - Safety Analysis Set (XX AEs in XX patients)

| = | 120 1222 | | | 2007 1 | 22242 020 04 | * (111111111 | | 22 51112 | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Cohort | Patient | Sex | Age | Date of | Number of | Adverse Event | | | | | | | | | | | | |
| | | Identification | | (years) | first dose | cycles | PT | Onset | End | Event | Date when | Intensity | Highest | AESI | irAE | IrAE | Tislelizu | mab | Outcome |
| | | Number | | | | received | | date | date | period | AE became | at onset | intensity | | (BG | accor | | | |
| | | Number | | | | received | | uute | date | period | | | interisity | | l | | Relation- | Action | |
| | | | | | | | | | | | serious | date | | | charte | ding | ship | taken | |
| | | | | | | | | | | | | | | | r) | to IC | Ship | taken | |
| Г | | X | Х | XX | XX/XX/XXXX | Х | XX | XX/XX/ | XX/XX/ | XX | XX/XX/XXXX | X | X | XX | XX | XX | X | XX | XX |
| | | | | | 7 - 7 | | | XXXX | XXXX | | , , | | | | | | | | |
| | | | | | | | | ^^^^ | | | | | | | | | | | |

<sup>\*</sup>Fatal AE are TEAE of grade 5

### 7.9.1.8 All AESI

### 7.9.1.8.1 Infusion-related reaction

Table 7.9-13 Description of infusion-related reaction by PT

| Preferred Term | Header | | |
|---------------------------|--------|---------|----|
| | Pá | Events | |
| Infusion-related reaction | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX |

### 7.9.1.8.2 Severe hypersensitivity reactions and flu-like symptoms

# Table 7.9-14 Description of severe hypersensitivity reactions and flu-like symptoms by PT

| Preferred Term | | Header | |
|---|---|---|---|
| | P | atients | Events |
| Severe hypersensitivity reactions and flu-like symptoms | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX |

# 7.9.1.8.3 Immune Related Aes (irAE) according to investigator

Table 7.9-15 Description of irAE according to investigator by PT

| Tuble 715 To Description of Hill according | <b>CO 121</b> ( CO | erent of a | |
|---|---|---|---|
| Type of AESI Preferred Term | | Header | |
| Treferred Term | Pa | Patients | |
| Immune-related adverse events according to | XX | (XX.X%) | XX |
| investigator | | | |
| PT1 | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX |

<u>Listing 7.9-2 All grade immune related Adverse Events according to investigator - Safety Analysis Set (XX AE reported by XX patients)</u>

| Coho | rt Patient | Sex | Age | Safety | Date of | Number | r Adverse Event | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Identification | | (yrs) | Analysis | first dose | of | irAE | PT | Onset | End date | Date | Intensity | Grade | Tislelizu | ımab | Outcome |
| | Number | | | Set | | cycles | according | | date | | when AE | at onset | | Relation- | Action | |
| | | | | | | received | to | | | | became | date | | ship | taken | |
| | | | | | | | Beigene | | | | serious | | | | | |
| | | | | | | | Charter | | | | | | | | | |
| X | XX | X | XX | XX | XX/XX/XXXX | X | X | XX | XX/XX/XXXX | XX/XX/XXXX | XX/XX/XXXX | X | X | X | XX | XX |

100 / 114

# 7.9.1.8.4 Immune Related AEs (irAE) according to Beigene charter

# 7.9.1.8.4.1 Grade ≥ 3

Table 7.9-16 Description of irAEs with grade >= 3 according to Beigene charter

| Type of | irAE | Header | | |
|-----------------------------|------|--------|---------|----|
| Preferred Term | İ | P | Events | |
| irAE with grade >= 3 | | XX | (XX.X%) | XX |
| Immune-mediated pneumonitis | | XX | (XX.X%) | XX |
| PT1 | | XX | (XX.X%) | XX |
| PT2 | | XX | (XX.X%) | XX |
| | | XX | (XX.X%) | XX |
| Immune-mediated pneumonitis | | XX | (XX.X%) | XX |
| PT1 | | XX | (XX.X%) | XX |
| PT2 | | XX | (XX.X%) | XX |
| | | XX | (XX.X%) | XX |
| | | XX | (XX.X%) | XX |
| PT1 | | XX | (XX.X%) | XX |
| PT2 | | XX | (XX.X%) | XX |
| l | | XX | (XX.X%) | XX |

Listing 7.9-3 Immune related Adverse Events with grade >= 3 - Safety Analysis Set (XX AE reported by XX patients)

| Coho | Patient | Se | Age | Safety | Date of | Numbe | | Adverse Event | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| rt | Identificati | x | (yrs | Analys | first | r of | irAE | PT | Onset | End date | Date | Intensit | Grad | Tislelizu | umab | Outcom |
| | on Number | | ) | is Set | dose | cycles | according | | date | | when AE | y at | e | Relatio | Actio | e |
| | | | | | | receive | to | | | | became | onset | | n-ship | n | |
| | | | | | | d | investigat | | | | serious | date | | • | take | |
| | | | | | | | or | | | | | | | | n | |
| V | XX | Х | XX | XX | XX/XX/XX | X | X | X | XX/XX/XX | XX/XX/XX | XX/XX/XX | X | Х | X | XX | XX |
| X | | _ ^ | | ^/^ | | | | | MyMyM | MyMym | MyMym | | | | ^/^ | /// |

# 7.9.1.9 All grade

Listing 7.9-4 All grade immune related Adverse Events according to Beigene charter - Safety Analysis Set (XX AE reported by XX patients)

| Coho | Patient | Se | Age | Safety | Date of | Numbe | Adverse Event | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| rt | Identificati | X | (yrs | Analys | first | r of | irAE | PT | Onset | End date | Date | Intensit | Grad | Tisleliz | umab | Outcom |
| | on Number | | ) | is Set | dose | cycles | according | | date | | when AE | y at | е | Relatio | Actio | e |
| | | | | | | receive | to | | | | became | onset | | n-ship | n | |
| | | | | | | d | investigat | | | | serious | date | | | take | |
| | | | | | | | or | | | | | | | | n | |
| X | XX | X | XX | XX | XX/XX/XX | X | X | X | XX/XX/XX | XX/XX/XX | XX/XX/XX | Х | X | X | XX | XX |
| | | | | | XX | | | X | XX | XX | XX | | | | | |

### 7.9.2 Serious Adverse Events

### 7.9.2.1 Summary

Table 7.9-17 Characteristics of Treatment Emergent Serious Adverse Events

| Table 7.7-17 Characteristics of 1. | tetter Line |
|--------------------------------------|-------------|
| | Header |
| TEAE onset Intensity | |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| 4 | XX (XX.X%) |
| 5 | XX (XX.X%) |
| TEAE highest Intensity | |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| 4 | XX (XX.X%) |
| 5 | XX (XX.X%) |
| Relationship with Tislelizumab | |
| Related | XX (XX.X%) |
| Unrelated | XX (XX.X%) |
| Action taken with Tislelizumab | |
| Permanent stop | XX (XX.X%) |
| Temporarily stop | XX (XX.X%) |
| Dose adaptation | XX (XX.X%) |
| Unchanged | XX (XX.X%) |
| Temporarily stop and Dose adaptation | XX (XX.X%) |
| Outcome | |
| Not recovered/Not resolved | XX (XX.X%) |
| Recovered/Resolved | XX (XX.X%) |
| Recovered/Resolved with sequelae | XX (XX.X%) |
| Death | XX (XX.X%) |
| Unknown | XX (XX.X%) |
| AESI | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

### 7.9.2.2 Treatment-emergent serious adverse events

Table 7.9-18 Description of treatment-emergent SAEs by SOC/PT

| System Organ Class | | Header | |
|------------------------|----|---------|--------|
| Preferred Term | P | atients | Events |
| Treatment-emergent SAE | XX | (XX.X%) | XX |
| SOC1 | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX |
| SOC2 | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX |

Table 7.9-19 Description of treatment-emergent SAEs by highest grade and SOC/PT - Cohort 1

| Table 7.5-17 Descr | tote 7.3-13 Description of treatment-emergent SAEs by mignest grade and SOC/1 1 - Conort 1 | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | | | | | Safet | y Analysis Set | - Cohort 1 | L | | | | | |
| Preferred Term | | | | | | | | N=XX | | | | | | | |
| | | Grade 1 | | | Grade 2 | | | Grade 3 | | | Grade 4 | | | Grade 5 | |
| İ | Pá | atients | Events | Pa | atients | Events | P | atients | Events | Pa | itients | Events | P | atients | Events |
| Treatment- | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| emergent SAE | | | | | | | | | | | | | | | |
| SOC1 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| SOC2 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |

# Table 7.9-20 Description of treatment-emergent SAEs by highest grade and SOC/PT - Cohort 2

<u>Listing 7.9-5 Treatment-emergent SAEs reported by patients - Safety Analysis Set (XX SAEs reported by XX patients)</u>

| C | Cohort | Patient | Sex | Age | | Number of | | | | Adver | se Event | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Identification | | (years) | Date of first | | | | | Date when AE | Intensity | Highest | Tislelizun | nab | Outcome |
| | | Number | | | dose | cycles | PT | Onset date | End date | became serious | at onset | intensity | Relationship | Action | |
| | | | | | | received | | | | | date | intensity | | taken | |
| | Χ | X | X | XX | XX/XX/XXXX | X | XX | XX/XX/XXXX | XX/XX/XXXX | XX/XX/XXXX | X | X | X | XX | XX |

7.9.2.3 Treatment-emergent SAEs leading to discontinuation of study treatment

<u>Table 7.9-21 Description of treatment-emergent SAEs leading to discontinuation of Tislelizumab by SOC/PT</u>

| System Organ Class<br>Preferred Term | | Header | |
|---|---|---|---|
| | F | Patients | |
| Treatment-emergent SAE leading to discontinuation of<br>Tislelizumab | XX | (XX.X%) | XX |
| SOC1 | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX |
| SOC2 | XX | (XX.X%) | XX |
| PT1 | XX | (XX.X%) | XX |
| PT2 | XX | (XX.X%) | XX |
| | XX | (XX.X%) | XX |

Table 7.9-22 Description of treatment-emergent SAEs leading to discontinuation of Tislelizumab by grade and SOC/PT - Cohort 1

| System Organ Class<br>Preferred Term | | Safety Analysis Set - Cohort 1<br>N=XX | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Grade | Grade 1 | | | | | Grade 3 | | Grade 4 | | | | Grade 5 | |
| | Patients | Events | F | atients | Events | | Patients | Events | P | Patients | Events | | Patients | Events |
| Treatment-emergent SAE | XX (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| leading to discontinuation of<br>Tislelizumab | | | | | | | | | | | | | | |
| SOC1 | XX (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT1 | XX (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT2 | XX (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| | XX (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| SOC2 | XX (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT1 | XX (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| PT2 | XX (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |
| | XX (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX | XX | (XX.X%) | XX |

Table 7.9-23 Description of treatment-emergent SAEs leading to discontinuation of Tislelizumab by grade and SOC/PT - Cohort 2

# 7.9.3 Second primary malignancies

Table 7.9-24 Description of other primary malignancies\* by SOC/PT

| System Organ Class<br>Preferred Term | Header | | | |
|---|---|---|---|---|
| Preferred Term | İ | P | Events | |
| Other malignancy | The state of the s | XX | (XX.X%) | XX |
| SOC1 | | XX | (XX.X%) | XX |
| PT1 | | XX | (XX.X%) | XX |
| PT2 | | XX | (XX.X%) | XX |
| | | XX | (XX.X%) | XX |
| SOC2 | | XX | (XX.X%) | XX |
| PT1 | 1 | XX | (XX.X%) | XX |
| PT2 | | XX | (XX.X%) | XX |
| | | XX | (XX.X%) | XX |

<sup>\*</sup> Per other primary malignancy page

Listing 7.9-6 Narratives of other primary malignancies - Safety Analysis Set (XX other

malignancies reported by XX patients)

| Cohort | Patient Identification<br>Number | Cohort | Date of first administration of<br>Tislelizumab | Date of<br>diagnosis | Narrative of other primary malignancy |
|---|---|---|---|---|---|
| X | X | X | XX/XX/XXXX | XX/XX/XXXX | XXXXX |

### 7.9.4 Deaths

Table 7.9-25 Deaths

| | Header |
|-------------------------------------------------|------------|
| Death | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, cause of death | |
| Lymphoma | XX (XX.X%) |
| Adverse event | XX (XX.X%) |
| Other reason | XX (XX.X%) |
| Unknown | XX (XX.X%) |
| If other cause, specification | |
| Toxicity of additional treatment | XX (XX.X%) |
| Unrelated cancer | XX (XX.X%) |
| Other concurrent illness | XX (XX.X%) |
| Other | XX (XX.X%) |
| If other reason, specification | |
| XXX | XX (XX.X%) |
| XXX | XX (XX.X%) |
| Death from cause other than disease progression | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Period of death | |
| Before treatment | XX (XX.X%) |
| During treatment | XX (XX.X%) |
| After treatment | XX (XX.X%) |

TIRHOL – Statistical Analysis Plan

Version 1.0 – 12APR2023

Table 7.9-26 Disease status at death

| | Header |
|-------------------------|------------|
| Disease status at death | |
| Complete Response | XX (XX,X%) |
| Partial Response | XX (XX,X%) |
| Stable Disease | xx (xx.x%) |
| Progressive Disease | XX (XX,X%) |
| Not Evaluated | xx (xx,x%) |
| Missing | xx (xx.x%) |

Listing 7.9-7 Deaths - Safety Analysis Set (XX patients)

| Cohort | Patient<br>Identification<br>Number | Sex | Age<br>(years) | Date of first<br>dose | Number<br>of cycles<br>received | Last administration | Study duration (months) | trea | nanent<br>tment<br>tinuation | Death within 90 days after discontinuation of study | De | eath |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | (Y/N) | Reason | treatment | Date | Cause |
| X | XXXX | Х | XX | XX/XX/XXXX | XX | XX/XX/XXXX | XX | XX | XX | X | XX/XX/XXXX | XX |

# Listing 7.9-8 Narratives of deaths due to SAE - Safety Analysis Set (XX patients)

| Cohort | Patient Identification Number | Narratives of fatal SAE |
|--------|-------------------------------|-------------------------|
| Х | XXXXXXXXXXXXX | Χ |

EN-SOP-ST-03-Temp-01-SAP Template (Phase II/III) – V2,0 - Effective date: 14/12/2016 107 / 114

### 7.9.5 Clinical Laboratory / Vital signs

7.9.5.1 Hematology

Table 7.9-27 Hematology: Shifts from baseline to worst post baseline grade - Cohort 1

| Hematology (Unit) | og , : omres ir om | Duscillic to Wol | Baseline | | | |
|---|---|---|---|---|---|---|
| CTCAE grade | Grade 0-1 | Grade 2 | Grade 3 | Grade 4 | Missing | Total |
| | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Hemoglobin (g/dL) - | 11 751 | 11 751 | 11 701 | 11 701 | 11 751 | 11 701 |
| low | | | | | | |
| Grade 0-1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | l xx | XX (XX.X%) |
| Grade 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Grade 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Grade 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Missing | XX | XX | XX | XX | XX | XX |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Platelet (G/L) | ΛΛ (ΛΛ.Λ /0) | ΛΛ (ΛΛ.Λ /0) | ΛΛ (ΛΛ.Λ /0) | ΛΛ (ΛΛ.Λ /0) | | ΛΛ (ΛΛ.Λ /0) |
| Grade 0-1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Grade 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Grade 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Grade 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Missing | XX (XX.X 70) | XX | XX (XX.X 70) | XX (XX.X 70) | XX | XX (XX.X 70) |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Absolute Neutrophil | AA (AA.A 70) | AA (AA.A70) | ΛΛ (ΛΛ.Λ <i>7</i> 0) | ΛΛ (ΛΛ.Λ 70) | | AA (AA.A 70) |
| Count (G/L) | | | | | | |
| Grade 0-1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Grade 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Grade 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Grade 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Missing | XX (XX.X 70) | XX | XX | XX (XX.X 70) | XX | XX |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Lymphocyte (G/L) - | AA (AA.A 70) | AA (AA.A 70) | AA (AA.A 70) | ΛΛ (ΛΛ.Λ /0) | | AA (AA.A 70) |
| low | | | | | | |
| Grade 0-1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Grade 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Grade 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Grade 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Missing | XX (XX.X-76) | XX | XX (XX.X-76) | XX (XX.X-70) | XX | XX (XX.X-76) |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Lymphocyte (G/L) - | ΛΛ (ΛΛ.Λ /0 <i>)</i> | λλ (λλ.λ /0) | ΛΛ (ΛΛ.Λ /0) | ΛΛ (ΛΛ.Λ /0) | ^^ | λλ (λλ.λ /0) |
| high | | | | | | |
| Grade 0-1 | NA | NA | NA | NA | NA | NA |
| Grade 0-1<br>Grade 2 | NA<br>NA | XX (XX.X%) | XX (XX.X%) | NA<br>NA | XX | XX (XX.X%) |
| Grade 2<br>Grade 3 | NA<br>NA | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%) | NA<br>NA | XX | XX (XX.X%) |
| Grade 4 | NA<br>NA | NA | NA (XX.X%) | NA<br>NA | NA NA | NA |
| Missing | NA<br>NA | XX | XX | NA<br>NA | XX | XX |
| Total | NA<br>NA | XX (XX.X%) | XX (XX.X%) | NA<br>NA | XX | XX (XX.X%) |
| TUM | NA | XX (XX.X%) | AA (AA.A%) | NA NA | | ۸۸ (۸۸.۸%) |

Only patients with at least one assessment (either baseline or postbaseline) were included in the table. The percentages were based on the number of patients with at least one assessment (either baseline or postbaseline).

Laboratory results were graded using NCI-CTCAE Version 5.

Hemoglobin - low: grade 0-1: >= 10.0 g/dL / grade 2: [8.0; 10.0 [g/dL] / grade 3: <8.0 g/dL

Platelet: grade 0-1: >=75.0 G/L / grade 2:  $[50.0; 75[.0 \text{ G/L / grade } 3: [25.0; 50.0] \text{ G/L / grade } 4: <25.0 \text{ G/$ 

Absolute Neutrophil Count: Grade0-1: >=1.5 G/L / grade 2: [1.0; 1.5] G/L / grade 3: [0.5; 1.0] G/L / grade 4: <0.5 G/L

Lymphocyte – low: grade 0-1: 0.8 >= G/L / grade 2: [0.5; 0.8[ G/L; grade 3: [0.2; 0.5[ G/L / grade 4: <0.2 G/L

Lymphocyte - high: grade 2: ]4; 20] G/L / grade 3: >20 G/L

<u>Table 7.9-28 Hematology: Shifts from baseline to worst post baseline grade - Cohort 2</u>
<u>Table 7.9-29 Hematology: Summary of Increase in 2 or More Grades as Compared with Baseline</u>

| - Conort 1 | | | | | | |
|---|---|---|---|---|---|---|
| Hematology (Unit) | Baseline | | | | | |
| CTCAE grade | Grade 0-1 | Grade 2 | Grade 3 | Grade 4 | Missing | Total |
| | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Hemoglobin (g/dL) - low | | | | | | |
| No increase or increase in one grade | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Increase in 2 or More Grades | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Platelet (G/L) | | | | | | |

| No increase or increase in one grade | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
|---|---|---|---|---|---|---|
| Increase in 2 or More Grades | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Absolute Neutrophil Count (G/L) | | | | | | |
| No increase or increase in one grade | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Increase in 2 or More Grades | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Lymphocyte (G/L) - low | | | | | | |
| No increase or increase in one grade | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Increase in 2 or More Grades | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Lymphocyte (G/L) - high | | | | | | |
| No increase or increase in one grade | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |
| Increase in 2 or More Grades | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X%) |

Only patients with at least one assessment (either baseline or postbaseline) were included in the table. The percentages were

based on the number of patients with at least one assessment (either baseline or postbaseline).

Laboratory results were graded using NCI-CTCAE Version 5.

Hemoglobin - low: grade 0-1: >= 10.0 g/dL / grade 2: [8.0; 10.0 [ g/dL / grade 3: < 8.0 g/dL )

Platelet: grade 0-1: >=75.0 G/L / grade 2: [50.0; 75[.0 G/L / grade 3: [25.0; 50.0[ G/L / grade 4: <25.0 G/L / grade 3: [25.0; 50.0] G/L / grade 4: <25.0 G/L

Absolute Neutrophil Count: Grade0-1: >=1.5 G/L / grade 2: [1.0; 1.5[ G/L / grade 3: [0.5; 1.0[ G/L / grade 4: <0.5 G/L

Lymphocyte - low: grade 0-1: 0.8 >= G/L / grade 2: [0.5; 0.8[ G/L; grade 3: [0.2; 0.5[ G/L / grade 4: <0.2 G/L ] ] ] ) | (0.2 in the context of the conte

Lymphocyte - high: grade 2: ]4; 20] G/L / grade 3: >20 G/L

<u>Table 7.9-30 Hematology: Summary of Increase in 2 or More Grades as Compared with Baseline - Cohort 2</u>

#### 7.9.5.2 Biochemistry

Table 7.9-31 Biochemistry: Shifts from baseline to worst post baseline grade - Cohort 1

| Biochemistry (Unit) | | | | Baseline | | | |
|---|---|---|---|---|---|---|---|
| CTCAE grade | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Missing | Total |
| | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| ALT (IU/L) | | | | | | | |
| Grade 0 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X9 |
| Grade 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X9 |
| Grade 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| AST (IU/L) | | | | | | | |
| Grade 0 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Total bilirubin | | | | | | | - |
| (µmol/L) | | | | | | | |
| Grade 0 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.X <sup>q</sup> |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Alkaline phosphatase | | | | | | | |
| (IU/L) | | | | | | | |
| Grade 0 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Serum creatinine | | | | | | | |
| (µmol/L) | | | | | | | |
| Grade 0 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Grade 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX | XX (XX.Xº |

Only patients with at least one assessment (either baseline or postbaseline) were included in the table. The percentages were based on the number of patients with at least one assessment (either baseline or postbaseline). Laboratory results were graded using NCI-CTCAE Version 5.0.

ALT - high: grade 1: ]ULN;  $3.0 \times ULN$ ] if baseline was normal; ]1.5 x baseline -  $3.0 \times Daseline$ ] if baseline was abnormal / grade 2: ]3.0 x ULN;  $5.0 \times ULN$ ] if baseline was normal; ]3.0 x baseline;  $5.0 \times Daseline$ ] if baseline was abnormal / grade 3: ]5.0 x ULN; 20.0 x ULN] if baseline was normal; ]5.0 x baseline; 20.0 x baseline] if baseline was abnormal / grade 4: >20.0 x ULN if baseline was normal; >20.0 x baseline if baseline was abnormal

AST - high: grade 1: ]ULN;  $3.0 \times ULN$ ] if baseline was normal; ]1.5 x baseline -  $3.0 \times Daseline$ ] if baseline was abnormal / grade 2: ]3.0 x ULN;  $5.0 \times ULN$ ] if baseline was normal; ]3.0 x baseline;  $5.0 \times Daseline$ ] if baseline was abnormal / grade 3: ]5.0 x ULN; 20.0 x ULN] if baseline was normal; ]5.0 x baseline; 20.0 x baseline] if baseline was abnormal / grade 4: >20.0 x ULN if baseline was normal; >20.0 x baseline if baseline was abnormal

Total bilirubin: grade 1: ]ULN; 1.5 x ULN] if baseline was normal; ]1.0 x baseline – 1.5 x baseline] if baseline was abnormal / grade 2: ]1.5 x ULN - 3.0 x ULN] if baseline was normal; ]1.5 x baseline - 3.0 x baseline] if baseline was abnormal / grade 3: ]3.0 x ULN - 10.0 x ULN] if baseline was normal; ]3.0 x baseline - 10.0 x baseline] if baseline was abnormal / grade 4: >10.0 x ULN if baseline was normal; >10 x baseline] if baseline was abnormal

Alkaline phosphatase: grade 1: ]ULN; 2.5 x ULN] if baseline was normal; ]2.0 x baseline – 2.5 x baseline] if baseline was abnormal / grade 2: ]2.5 x ULN - 5.0 x ULN] if baseline was normal; ]2.5 x baseline - 5.0 x baseline] if baseline was abnormal /

grade 3: ]5.0 x ULN - 20.0 x ULN] if baseline was normal; ]5.0 x baseline - 20.0 x baseline] if baseline was abnormal / grade 4: >20.0 x ULN if baseline was normal; >20 x baseline] if baseline was abnormal

Serum creatinine: grade 1: ]ULN; 1.5 x ULN] / grade 2: ]1.5 x ULN - 3.0 x ULN] / grade 3: ]3.0 x ULN - 6.0 x ULN] / grade 4: >6.0 x ULN

#### Table 7.9-32 Biochemistry: Shifts from baseline to worst post baseline grade - Cohort 2

Table 7.9-33 Biochemistry: Summary of Increase in 2 or More Grades as Compared with Baseline

| <u>- Cohort 1</u> | | | | | | | |
|---|---|---|---|---|---|---|---|
| Biochemistry (Unit) | | | | Baseline | | | |
| CTCAE grade | Grade 0<br>N=XX | Grade 1<br>N=XX | Grade 2<br>N=XX | Grade 3<br>N=XX | Grade 4<br>N=XX | Missing<br>N=XX | Total<br>N=XX |
| ALT (IU/L) | | | | | | | |
| No increase or increase in one | XX | XX | XX | XX | XX | XX | XX |
| grade | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | | (XX.X%) |
| Increase in 2 or More Grades | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | | (XX.X%) |
| AST (IU/L) | | | | | | | |
| No increase or increase in one | XX | XX | XX | XX | XX | XX | XX |
| grade | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | | (XX.X%) |
| Increase in 2 or More Grades | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | | (XX.X%) |
| Total bilirubin (µmol/L) | | | | | | | |
| No increase or increase in one | XX | XX | XX | XX | XX | XX | XX |
| grade | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | | (XX.X%) |
| Increase in 2 or More Grades | XX | XX | XX | XX | XX | XX | XX |
| -11 12 1 1 1 1 1 1 1 1 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | - | (XX.X%) |
| Alkaline phosphatase (IU/L) | | | | | | | |
| No increase or increase in one | XX | XX | XX | XX | XX | XX | XX |
| grade | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | | (XX.X%) |
| Increase in 2 or More Grades | XX | XX | XX | XX | XX | XX | XX |
| 6 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | | (XX.X%) |
| Serum creatinine (µmol/L) | VV | VV | VV | VV | VV | | W |
| No increase or increase in one | XX | XX | XX | XX | XX | XX | XX |
| grade | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | \ \vv | (XX.X%) |
| Increase in 2 or More Grades | XX | XX | XX | XX | XX | XX | XX<br>(XX.X%) |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | | (٨٨.٨%) |

Only patients with at least one assessment (either baseline or postbaseline) were included in the table. The percentages were based on the number of patients with at least one assessment (either baseline or postbaseline). Laboratory results were graded using NCI-CTCAE Version 5.0.

ALT - high: grade 1: ]ULN; 3.0 x ULN] if baseline was normal; ]1.5 x baseline - 3.0 x baseline] if baseline was abnormal / grade 2: ]3.0 x ULN; 5.0 x ULN] if baseline was normal; ]3.0 x baseline; 5.0 x baseline] if baseline was abnormal / grade 3: ]5.0 x ULN; 20.0 x ULN] if baseline was normal; ]5.0 x baseline; 20.0 x baseline] if baseline was abnormal / grade 4: >20.0 x ULN if baseline was normal; >20.0 x baseline if baseline was abnormal

AST - high: grade 1: ]ULN;  $3.0 \times ULN$ ] if baseline was normal; ]1.5 x baseline -  $3.0 \times DLN$  if baseline was abnormal / grade 2: ]3.0 x ULN;  $5.0 \times ULN$ ] if baseline was normal; ]3.0 x baseline;  $5.0 \times DLN$  if baseline was abnormal / grade 3: ]5.0 x ULN; 20.0 x ULN] if baseline was normal; ]5.0 x baseline; 20.0 x baseline] if baseline was abnormal / grade 4: >20.0 x ULN if baseline was normal; >20.0 x baseline if baseline was abnormal

Total bilirubin: grade 1: ]ULN; 1.5 x ULN] if baseline was normal; ]1.0 x baseline – 1.5 x baseline] if baseline was abnormal / grade 2: ]1.5 x ULN - 3.0 x ULN] if baseline was normal; ]1.5 x baseline - 3.0 x baseline] if baseline was abnormal / grade 3: ]3.0 x ULN - 10.0 x ULN] if baseline was normal; ]3.0 x baseline - 10.0 x baseline] if baseline was abnormal / grade 4: >10.0 x ULN if baseline was normal; >10 x baseline] if baseline was abnormal

Alkaline phosphatase: grade 1: ]ULN; 2.5 x ULN] if baseline was normal; ]2.0 x baseline – 2.5 x baseline] if baseline was abnormal / grade 2: ]2.5 x ULN - 5.0 x ULN] if baseline was normal; ]2.5 x baseline - 5.0 x baseline] if baseline was abnormal / grade 3: ]5.0 x ULN - 20.0 x ULN] if baseline was normal; ]5.0 x baseline - 20.0 x baseline] if baseline was abnormal / grade 4: >20.0 x ULN if baseline was normal; >20 x baseline] if baseline was abnormal

Serum creatinine: grade 1: ]ULN;  $1.5 \times ULN$ ] / grade 2: ] $1.5 \times ULN - 3.0 \times ULN$ ] / grade 3: ] $3.0 \times ULN - 6.0 \times ULN$ ] / grade 4: >6.0 x ULN

# <u>Table 7.9-34 Biochemistry: Summary of Increase in 2 or More Grades as Compared with Baseline - Cohort 2</u>

### 7.9.5.3 Vital sign

Table 7.9-35 Vital signs during treatment

| Vital sign examination performed at | |
|-------------------------------------|-------------|
| g caumination periorited at | |
| cycle 1 | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Systolic blood pressure (mmHG) | |
| N | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Diastolic blood pressure (mmHG) | |
| N | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Pulse (beats/min) | |
| N | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Body temperature (°C) | |
| N | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |

# 7.9.6 Pregnancies

# Listing 7.9-9 Narratives of pregnancies - Safety Analysis Set (XX patients)

| Cohort | Patient Identification Number | Narratives of pregnancies |
|--------|-------------------------------|---------------------------|
| X | XXXXXXXXXXXXX | X |

### 7.10 Prior and concomitant treatments

### 7.10.1 Prior treatments reported at enrollment

Table 7.10-1 Corticosteroids treatments reported at enrollment

| | Header |
|---------------------------------------------------|------------|
| Corticosteroids treatments reported at enrollment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, still ongoing | |
| No | XX (XX.X%) |
| yes | XX (XX.X%) |
| ATC4 | |
| | XX (XX.X%) |
| | XX (XX.X%) |
| Indication | |
| | XX (XX.X%) |
| | XX (XX.X%) |

Note: A patient with multiple occurrences of the same concomitant treatment is counted only once

Table 7.10-2 Prior treatments reported at enrollment

| | Header |
|-----------------------------------------------|------------|
| Concomitant treatments reported at enrollment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, still ongoing | |
| No | XX (XX.X%) |
| yes | XX (XX.X%) |
| ATC4 | |
| | XX (XX.X%) |
| | XX (XX.X%) |
| Indication | |
| *** | XX (XX.X%) |
| | XX (XX.X%) |

Note: A patient with multiple occurrences of the same concomitant treatment is counted only once

#### 7.10.2 Concomitant treatments

**Table 7.10-3 Concomitant treatments** 

| | Header |
|------------------------------------------------------|------------|
| Patients with at least one new concomitant treatment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, related to AE | |
| No . | XX (XX.X%) |
| yes | XX (XX.X%) |
| ATC4 | |
| | XX (XX.X%) |
| | XX (XX.X%) |
| Indication | |
| | XX (XX.X%) |
| | XX (XX.X%) |

Note: A patient with multiple occurrences of the same concomitant treatment is counted only once

Listing 7.10-1 Concomitant treatments - Safety Analysis Set (XX AEs in XX patients)

| Ī | Cohort | Patient | Sex | Age | Date of | Number | New concomitant treatment | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Identificati<br>on Number | | (years | first dose | of cycles<br>received | Drug<br>name<br>(INN) | Indication | Route | Start<br>date | ongoing | If not<br>ongoing,<br>end date | Related to<br>AE |
| | X | X | X | XX | XX/XX/XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | | | l | XX | | | | | | | | |